CLINICAL TRIAL: NCT04001803
Title: A Qualitative Hybrid III Implementation Study to Identify and Evaluate Strategies for Successful Implementation of the Cabotegravir + Rilpivirine Long-acting Injectable Regimen in the US
Brief Title: Study to Identify and Determine Best Implementation Practices for Injectable Cabotegravir+Rilpivirine in the United States (US)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 209493
Record Dates: First submitted 2019-06-10; First posted 2019-06-28 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections
Keywords: Antiretroviral therapy, HIV infections, cabotegravir, rilpivirine, long-acting intramuscular injection,
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with HIV infection (Experimental): HIV-infected subjects receiving CAB LA+RPV LA will be included in this arm.
  Interventions: Drug: CAB LA+RPV LA

INTERVENTIONS:
Drug: CAB LA+RPV LA — Subjects will receive one tablet of CAB 30 milligram(mg) + RPV 25 mg once daily from Day 1 for 1 month. During month 1, subjects will receive 600 mg of CAB LA injection+ 900 mg of RPV LA injection. Following Month 1, subjects will receive 400mg of CAB LA + 600mg of RPV LA at each subsequent injection.

SUMMARY:
Chronic human immunodeficiency virus (HIV) infection in adults continues to be characterized by increased development of resistant virus, increased transmission of resistant virus and issues associated with the long-term toxicity of anti-retroviral therapy (ART), despite advances in development of new ART, which provides extensive insight in management of HIV-infected individuals. Cabotegravir (CAB) is a potent integrase inhibitor (INI) and rilpivirine (RPV) is a potent non-nucleoside reverse transcriptase inhibitor (NNRTI). A two-drug regimen (DR)with CAB plus RPV long acting (LA) product offers many potential advantages over daily oral regimens including better tolerability, improved compliance, adherence, less likely to develop resistance, and overall treatment satisfaction in virologically suppressed subjects. This is a single-arm, open-label, multicenter, short term facilitation study to evaluate the effect of an implementation strategy on the degree of acceptability, appropriateness, feasibility, fidelity and sustainability of clinical practices to deliver the CAB+RPV LA regimen to HIV infected subjects and to also measure subject satisfaction by recording timeliness of visits, length of visit and their education. Approximately 135 subjects will be enrolled in the study and the total duration of the study will be approximately 52-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand and comply with protocol requirements, instructions, and restrictions;
* Understand the long-term commitment to the study and be likely to complete the study as planned;
* Be considered appropriate candidates for participation in an investigative clinical trial with oral and intramuscularly injectable medications (e.g., no active substance use disorder, acute major organ disease, or planned long-term work assignments out of the country, etc.).

All Participants eligible for enrolment in the study must meet all of the following criteria:

* Aged 18 years or older at the time of signing the informed consent.
* HIV-1 infected and must be on an active highly active antiretroviral therapy (HAART) (2 or 3 drug) regimen for at least 6 months prior to Screening. Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability/safety, access to medications, or convenience/simplification, and must NOT have been done for treatment failure (HIV-1 RNA >=200 c/mL).

Acceptable stable ARV regimens prior to Screening include 2 NRTIs plus:

• INI (either the initial or second Combination antiretroviral therapy (cART) regimen)

* NNRTI (either the initial or second cART regimen)
* Boosted prediction interval (PI) (or atazanavir [ATV] unboosted) (must be either the initial cART regimen or one historical within class switch is permitted due to safety/tolerability)
* Any suppressed participants on a triple ART regimen for at least 6 months who had their regimen switched to a 2DR of dolutegravir (DTG)/RPV

  - Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: at least one within 6 months prior to Screening;
  * Plasma HIV-1 RNA <50 c/mL at Screening;
  * A female participant is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin (hCG) test at screen and at Day 1), not lactating, and at least one of the following conditions applies:

    1. Non-reproductive potential defined as:
* Pre-menopausal females with one of the following:

  * Documented tubal ligation
  * Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
  * Hysterectomy
  * Documented Bilateral Oophorectomy
* Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

  b. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, and for at least 30 days after discontinuation of all oral study medications and for at least 52 weeks after discontinuation of CAB LA and RPV LA. The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception.

  - Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol. Eligible participants or their legal guardians (and next of kin when locally required), must sign a written Informed Consent Form before any protocol-specified assessments are conducted. Enrolment of participants who are unable to provide direct informed consent is optional and will be based on local legal/regulatory requirements and site feasibility to conduct protocol procedures.

Exclusion Criteria:

* Within 6 months prior to Screening, plasma HIV-1 RNA measurement >=50 c/mL;
* During the previous 12 months, any confirmed HIV-1 RNA measurement >=200 c/mL Exclusionary medical conditions
* Women who are pregnant, breastfeeding, or plan to become pregnant or breastfeed during the study
* Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy, and Cluster of Differentiation (CD4+) counts <200 cells/microliter are not exclusionary
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low.
* Participants who, in the investigator's judgment, pose a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* The participant has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV Deoxyribonucleic acid (DNA) as follows:

  * Participants positive for HBsAg are excluded;
  * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded Note: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.
* Participants who are anticipated to require HCV treatment within 12 months must be excluded. Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded; investigators must carefully assess if therapy specific for HCV infection is required. (HCV treatment on study may be permitted, following consultation and approval of the direct acting antiviral (DAA) drug based therapy being considered with the medical monitor).
* Participants with HCV co-infection will be allowed entry into this study if:

  * Liver enzymes meet entry criteria
  * HCV Disease has undergone appropriate work-up, and is not advanced. Additional information (where available) on participants with HCV coinfection at screening should include results from any liver biopsy, Fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment.
  * In the event that recent biopsy or imaging data is not available or inconclusive, the Fib-4 score will be used to verify eligibility

    * Fib-4 score >3.25 is exclusionary
    * Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation Fibrosis 4 Score Formula: (Age x AST) / (Platelets x ( sqr [ ALT ])
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis.
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to inclusion.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class.
* Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (<=325 milligram (mg) per day) or hereditary coagulation and platelet disorders such as haemophilia or Von Willebrand Disease.
* Corrected QT interval (QTc [Bazett]) >450 milli second (msec) or QTc (Bazett) >480 msec for subjects with bundle branch block). Exclusionary Laboratory Values or Clinical Assessments (a single repeat to determine eligibility is allowed).
* Any evidence of primary resistance based on the presence of any major known INI or NNRTI resistance-associated mutation, except for K103N, (International acquired immune deficiency syndrome [AIDS] Society [IAS]-USA) by any historical resistance test result.
* ALT >=5 × Upper Limit Normal (ULN) or ALT >=3xULN and bilirubin >=1.5xULN (with >35% direct bilirubin) over the last 6 months.
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening phase to verify a result.
* Participant has estimated creatinine clearance <50 mL/min/1.73meter^2 via the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

Concomitant Medications

* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study;
* Treatment with any of the following agents within 28 days of Day 1:

  * radiation therapy;
  * cytotoxic chemotherapeutic agents;
  * tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid [INH]);
  * anti-coagulation agents;
  * Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons. Note: Participants using short-term (e.g. <=21 days) systemic corticosteroid treatment; topical, inhaled and intranasal corticosteroids are eligible for enrolment.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Use of medications which are associated with Torsade de Pointes must be discussed with the Medical Monitor to determine eligibility.
* Subjects receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication. Note: Any prohibited medications that decrease CAB or RPV concentrations should be discontinued for a minimum of four weeks or a minimum of three half-lives (whichever is longer) prior to the first dose and any other prohibited medications should be discontinued for a minimum of two weeks or a minimum of three half-lives (whichever is longer) prior to the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (9):
- United States (9):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on ViiV's data sharing criteria can be found at: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/

REFERENCES:
- [Background] Czarnogorski M, Garris CP, Dalessandro M, D'Amico R, Nwafor T, Williams W, Merrill D, Wang Y, Stassek L, Wohlfeiler MB, Sinclair GI, Mena LA, Thedinger B, Flamm JA, Benson P, Spreen WR. Perspectives of healthcare providers on implementation of long-acting cabotegravir plus rilpivirine in US healthcare settings from a Hybrid III Implementation-effectiveness study (CUSTOMIZE). J Int AIDS Soc. 2022 Sep;25(9):e26003. doi: 10.1002/jia2.26003. PMID 36094142
- [Derived] Garris CP, Czarnogorski M, Dalessandro M, D'Amico R, Nwafor T, Williams W, Merrill D, Wang Y, Stassek L, Wohlfeiler MB, Sinclair GI, Mena LA, Thedinger B, Flamm JA, Benson P, Spreen WR. Perspectives of people living with HIV-1 on implementation of long-acting cabotegravir plus rilpivirine in US healthcare settings: results from the CUSTOMIZE hybrid III implementation-effectiveness study. J Int AIDS Soc. 2022 Sep;25(9):e26006. doi: 10.1002/jia2.26006. PMID 36097674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 115 participants were enrolled in study and received study treatment. The 24 study staff population(HIV care providers,nurses/staff performing CAB+LA injections administrators/clinic managers)is not considered participants in the study and were not counted in the enrollment number nor reported in any modules that are considered for enrolled participants as study staff didn't have to complete the informed consent process and did not receive oral lead-in medication or CAB+RPV LA injections.
Pre-assignment Details: Study staff participants only provided input through the completion of surveys, semi-structured interviews and facilitation calls. Participant flow, Baseline characteristics or adverse events for study staff participants were not collected because it was not required per study design.
Groups:
- Participants With HIV Infection: In the Intervention Phase, participants with Human immunodeficiency virus (HIV) infection received one tablet of Cabotegravir (CAB) 30 milligrams (mg) + Rilpivirine (RPV) 25 mg once daily from Day 1 for 1 month. During Month 1, participants were administered 600 mg of CAB long-acting (LA) + 900 mg of RPV LA via intramuscular (IM) route. From Month 2, participants received 400 mg of CAB LA + 600 mg of RPV LA via IM route every month until Month 12. Participants continued CAB LA + RPV LA IM injection from Month 13 in the Extension Phase until it is commercially available. Participants were followed up for an additional 52 weeks if they discontinue the study treatment (after receiving at least 1 dose of CAB LA and /or RPV LA) and have started an alternative antiretroviral therapy (ART).
Period: Intervention Phase (Up to Month 12)
Arm/Group | Participants With HIV Infection
Started | 115
Completed | 102
Not Completed | 13
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 4
Period: Extension Phase (From Months 13 to 30)
Arm/Group | Participants With HIV Infection
Started | 101 (1 participant completed Intervention Phase but did not enter the Extension Phase (Participant Relocated))
Completed | 95
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Period: Long-term Follow-up Phase(Up to Week 52)
Arm/Group | Participants With HIV Infection
Started | 10 (85 participants who completed the Extension Phase did not enter Long-term follow-up Phase as they transitioned off CAB LA + RPV LA regimen to commercial available CAB LA + RPV LA.)
Completed | 7
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for Safety Population(comprised of all participants enrolled,who received atleast 1 dose of CAB LA+RPV LA).Study staff participants only provided input through completion of surveys,semi-structured interviews,facilitation calls and didn't have to complete the informed consent process and did not receive oral lead-in medication or CAB+RPV LA injections. Demographics for study staff participants were not collected because it was not required per study design
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan native | 5
  Black or African American | 42
  White-White/Caucasian/European heritage | 66
  Black or African American and White | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Acceptability of Intervention Measure (AIM) Total Score in Staff Study Participants at Month 4
Description: AIM is a four item survey that assessed the acceptability of an implementation process. The staff study participants were asked to indicate how much they agreed or disagreed with each of the 4 items in the AIM based on their current experiences with implementing the CAB + RPV injection treatment on a five point rating scale (1=completely disagree to 5=completely agree). The AIM total score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and Month 4
Population: All Staff study participants Population comprised of HIV care providers (HCPs), nurses/staff performing CAB+RPV LA injections and administrators/clinic managers at each investigational site.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Staff Study Participants: Staff study participants included HIV care providers (HCPs), nurses/staff performing CAB + RPV LA injections, and administrators/clinic managers at each investigational site. They provided input through the use of surveys, semistructured interviews (SSI) and via monthly facilitation calls
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 24
Scores on a scale | 0.00 (0.42)

2. Primary Outcome: Change From Baseline in AIM Total Score in Staff Study Participants at Month 12
Description: as for outcome 1
Time Frame: Baseline and Month 12
Population: All staff study participants population. Only those staff study participants who completed the survey were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 23
Scores on a scale | 0.02 (0.52)

3. Primary Outcome: Change From Baseline in AIM Total Score in Participants With HIV Infection at Month 4
Description: AIM is a four item survey that assessed the acceptability of an implementation process. The participants were asked about their impressions of the CAB LA + RPV LA injection treatment for treating HIV on a five point rating scale (1=completely disagree to 5=completely agree). The AIM total score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and Month 4
Population: Safety population consisted of all participants who were enrolled and received atleast one dose of CAB LA + RPV LA. Only those participants who completed the survey were included in the analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 105
Scores on a scale | 0.03 (0.74)

4. Primary Outcome: Change From Baseline in AIM Total Score in Participants With HIV Infection at Month 12
Description: as for outcome 3
Time Frame: Baseline and Month 12
Population: Safety population. Only those participants who completed the survey were included in the analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Scores on a scale | 0.19 (0.52)

5. Primary Outcome: Change From Baseline in Intervention Appropriateness Measure (IAM) Score in Staff Study Participants at Month 4
Description: IAM is a four item survey that assessed the appropriateness of an implementation process. The staff study participants were asked to indicate how much they agreed or disagreed with each of the 4 items in the IAM based on their current experiences with implementing the CAB + RPV injection treatment on a five point rating scale (1=completely disagree to 5=completely agree). The IAM total score ranges from 1 to 5 with 1 indicating the least appropriateness and 5 the most appropriateness. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and Month 4
Population: All Staff study participants population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 24
Scores on a scale | -0.03 (0.50)

6. Primary Outcome: Change From Baseline in IAM Score in Staff Study Participants at Month 12
Description: as for outcome 5
Time Frame: Baseline and Month 12
Population: All Staff study participant population. Only those staff study participants who completed the survey were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 23
Scores on a scale | 0.10 (0.43)

7. Primary Outcome: Change From Baseline in IAM Score in Participants With HIV Infection at Month 4
Description: IAM is a four item survey that assessed the appropriateness of an implementation process. The participants were asked to indicate how much they agreed or disagreed with each of the 4 items in the IAM based on their current experiences with implementing the CAB + RPV injection treatment on a five point rating scale (1=completely disagree to 5=completely agree). The IAM total score ranges from 1 to 5 with 1 indicating the least appropriateness and 5 the most appropriateness. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and Month 4
Population: Safety population. Only those participants who completed the survey were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 105
Scores on a scale | 0.05 (0.78)

8. Primary Outcome: Change From Baseline in IAM Score in Participants With HIV Infection at Month 12
Description: as for outcome 7
Time Frame: Baseline and Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Scores on a scale | 0.19 (0.58)

9. Primary Outcome: Change From Baseline in Feasibility of Intervention Measure (FIM) Total Score in Staff Study Participants at Month 4
Description: FIM is a four item survey that assessed the feasibility of an implementation process. The staff study participants were asked to indicate how much they agreed or disagreed with each of the 4 items in the FIM based on their current experiences with implementing the CAB + RPV injection treatment on a five point rating scale (1=completely disagree to 5=completely agree). The FIM total score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and Month 4
Population: All staff study participants Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 24
Scores on a scale | -0.02 (0.63)

10. Primary Outcome: Change From Baseline for FIM Total Score in Staff Study Participants at Month 12
Description: as for outcome 9
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 23
Scores on a scale | 0.07 (0.69)

11. Secondary Outcome: Number of Staff Study Participants Reported Helpfulness of Toolkit Resources at Month 4
Description: The helpfulness of the toolkit resources was identified using a 19-item survey and the helpfulness of the resources were rated on a five point scale where 1=Extremely helpful (EH), 2=Very helpful (VH), 3=Somewhat helpful (SH), 4=A little helpful (ALH) and 5=Not at all helpful (NAAH). Not Applicable (NA) in the categories mean response was not offered. The toolkit resources consisted of website for clinical staff, video on giving CAB + RPV LA, how to use new packaging card, study factsheet for healthcare providers, consultation aid, reminder e-application, reminder SMS/text, face-to-face training by healthcare staff, facilitation group calls, web-based (WB) treatment planner, WB health clinic capacity planning tool, injection flashcards, website for participants, what to expect factsheet, handbook, FAQ chatbot, trial guide app, video-what to expect and hot and cold packs. The number of participants with the rating on helpfulness for each toolkit resources at Month 4 is presented.
Time Frame: At Month 4
Population: All staff study participants population.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 24
Participants
  Website for clinical staff, EH | 2
  Website for clinical staff, VH | 3
  Website for clinical staff, SH | 3
  Website for clinical staff, ALH | 5
  Website for clinical staff, NAAH | 1
  Website for clinical staff, NA | 10
  Video on giving CAB + RPV LA injection, EH | 3
  Video on giving CAB + RPV LA injection, VH | 6
  Video on giving CAB + RPV LA injection, SH | 4
  Video on giving CAB + RPV LA injection, ALH | 2
  Video on giving CAB + RPV LA injection, NAAH | 0
  Video on giving CAB + RPV LA injection, NA | 9
  How to use new packaging card, EH | 0
  How to use new packaging card, VH | 6
  How to use new packaging card, SH | 3
  How to use new packaging card, ALH | 3
  How to use new packaging card, NAAH | 1
  How to use new packaging card, NA | 11
  Study factsheet for healthcare providers, EH | 1
  Study factsheet for healthcare providers, VH | 4
  Study factsheet for healthcare providers, SH | 8
  Study factsheet for healthcare providers, ALH | 1
  Study factsheet for healthcare providers, NAAH | 1
  Study factsheet for healthcare providers, NA | 9
  Consultation aid, EH | 0
  Consultation aid, VH | 4
  Consultation aid, SH | 4
  Consultation aid, ALH | 2
  Consultation aid, NAAH | 1
  Consultation aid, NA | 13
  Reminder-electronic (e)-application (app), EH | 1
  Reminder e-app, VH | 2
  Reminder e-app, SH | 1
  Reminder e-app, ALH | 2
  Reminder e-app, NAAH | 0
  Reminder e-app, NA | 18
  Reminder short message service (SMS)/text, EH | 1
  Reminder SMS/text, VH | 1
  Reminder SMS/text, SH | 1
  Reminder SMS/text, ALH | 2
  Reminder SMS/text, NAAH | 0
  Reminder SMS/text, NA | 19
  Face to face (F2F) training by healthcare staff, EH | 5
  F2F training by healthcare staff, VH | 6
  F2F training by healthcare staff, SH | 3
  F2F training by healthcare staff, ALH | 1
  F2F training by healthcare staff, NAAH | 0
  F2F training by healthcare staff, NA | 9
  Facilitation group calls, EH | 0
  Facilitation group calls, VH | 0
  Facilitation group calls, SH | 7
  Facilitation group calls, ALH | 8
  Facilitation group calls, NAAH | 4
  Facilitation group calls, NA | 5
  Web-based (WB) treatment planner, EH | 4
  WB treatment planner, VH | 5
  WB treatment planner, SH | 1
  WB treatment planner, ALH | 1
  WB treatment planner, NAAH | 1
  WB treatment planner, NA | 12
  WB health clinic capacity planning tool, EH | 0
  WB health clinic capacity planning tool, VH | 1
  WB health clinic capacity planning tool, SH | 0
  WB health clinic capacity planning tool, ALH | 0
  WB health clinic capacity planning tool, NAAH | 1
  WB health clinic capacity planning tool, NA | 22
  Injection flashcard for participants, EH | 2
  Injection flashcard for participants, VH | 2
  Injection flashcard for participants, SH | 5
  Injection flashcard for participants, ALH | 3
  Injection flashcard for participants, NAAH | 0
  Injection flashcard for participants, NA | 12
  Website for participants, EH | 0
  Website for participants, VH | 3
  Website for participants, SH | 4
  Website for participants, ALH | 2
  Website for participants, NAAH | 0
  Website for participants, NA | 15
  What to expect factsheet for participants, EH | 1
  What to expect factsheet for participants, VH | 5
  What to expect factsheet for participants, SH | 7
  What to expect factsheet for participants, ALH | 2
  What to expect factsheet for participants, NAAH | 0
  What to expect factsheet for participants, NA | 9
  Participant handbook, EH | 3
  Participant handbook, VH | 3
  Participant handbook, SH | 5
  Participant handbook, ALH | 0
  Participant handbook, NAAH | 1
  Participant handbook, NA | 12
  Frequently asked questions (FAQs) chatbot, EH | 0
  FAQs chatbot, VH | 1
  FAQs chatbot, SH | 3
  FAQs chatbot, ALH | 1
  FAQs chatbot, NAAH | 1
  FAQs chatbot, NA | 18
  Trial guide app, EH | 0
  Trial guide app, VH | 1
  Trial guide app, SH | 2
  Trial guide app, ALH | 1
  Trial guide app, NAAH | 1
  Trial guide app, NA | 19
  Video-what to expect, EH | 7
  Video-what to expect, VH | 4
  Video-what to expect, SH | 1
  Video-what to expect, ALH | 3
  Video-what to expect, NAAH | 1
  Video-what to expect, NA | 8
  Hot and cold packs for participants, EH | 5
  Hot and cold packs for participants, VH | 5
  Hot and cold packs for participants, SH | 6
  Hot and cold packs for participants, ALH | 2
  Hot and cold packs for participants, NAAH | 0
  Hot and cold packs for participants, NA | 6

12. Secondary Outcome: Number of Staff Study Participants Reported Helpfulness of Toolkit Resources at Month 12
Description: The helpfulness of the toolkit resources was identified using a 19-item survey and the helpfulness of the resources were rated on a five point scale where 1=Extremely helpful (EH), 2=Very helpful (VH), 3=Somewhat helpful (SH), 4=A little helpful (ALH) and 5=Not at all helpful (NAAH). Not Applicable (NA) in the categories mean response was not offered. The toolkit resources consisted of website for clinical staff, video on giving CAB + RPV LA, how to use new packaging card, study factsheet for healthcare providers, consultation aid, reminder e-application, reminder SMS/text, face-to-face training by healthcare staff, facilitation group calls, WB treatment planner, WB health clinic capacity planning tool, injection flashcards, website for participants, what to expect factsheet for participants, handbook, FAQ chatbot, trial guide app, video-what to expect and hot and cold packs. The number of participants with the rating on helpfulness for each toolkit resources at Month 12 is presented.
Time Frame: At Month 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 23
Participants
  Website for clinical staff, EH | 2
  Website for clinical staff, VH | 2
  Website for clinical staff, SH | 6
  Website for clinical staff, ALH | 0
  Website for clinical staff, NAAH | 0
  Website for clinical staff, NA | 13
  Video on giving CAB + RPV LA injection, EH | 4
  Video on giving CAB + RPV LA injection, VH | 6
  Video on giving CAB + RPV LA injection, SH | 7
  Video on giving CAB + RPV LA injection, ALH | 0
  Video on giving CAB + RPV LA injection, NAAH | 0
  Video on giving CAB + RPV LA injection, NA | 6
  How to use new packaging card, EH | 1
  How to use new packaging card, VH | 3
  How to use new packaging card, SH | 5
  How to use new packaging card, ALH | 0
  How to use new packaging card, NAAH | 0
  How to use new packaging card, NA | 14
  Study factsheet for healthcare providers, EH | 1
  Study factsheet for healthcare providers, VH | 6
  Study factsheet for healthcare providers, SH | 4
  Study factsheet for healthcare providers, ALH | 1
  Study factsheet for healthcare providers, NAAH | 0
  Study factsheet for healthcare providers, NA | 11
  Consultation aid, EH | 1
  Consultation aid, VH | 1
  Consultation aid, SH | 2
  Consultation aid, ALH | 5
  Consultation aid, NAAH | 0
  Consultation aid, NA | 14
  Reminder e-app, EH | 0
  Reminder e-app, VH | 1
  Reminder e-app, SH | 0
  Reminder e-app, ALH | 0
  Reminder e-app, NAAH | 1
  Reminder e-app, NA | 21
  Reminder SMS/text, EH | 1
  Reminder SMS/text, VH | 1
  Reminder SMS/text, SH | 0
  Reminder SMS/text, ALH | 1
  Reminder SMS/text, NAAH | 2
  Reminder SMS/text, NA | 18
  F2F training by healthcare staff, EH | 6
  F2F training by healthcare staff, VH | 10
  F2F training by healthcare staff, SH | 3
  F2F training by healthcare staff, ALH | 0
  F2F training by healthcare staff, NAAH | 0
  F2F training by healthcare staff, NA | 4
  Facilitation group calls, EH | 1
  Facilitation group calls, VH | 1
  Facilitation group calls, SH | 5
  Facilitation group calls, ALH | 5
  Facilitation group calls, NAAH | 4
  Facilitation group calls, NA | 7
  WB treatment planner, EH | 4
  WB treatment planner, VH | 1
  WB treatment planner, SH | 4
  WB treatment planner, ALH | 0
  WB treatment planner, NAAH | 1
  WB treatment planner, NA | 13
  WB health clinic capacity planning tool, EH | 0
  WB health clinic capacity planning tool, VH | 0
  WB health clinic capacity planning tool, SH | 2
  WB health clinic capacity planning tool, ALH | 1
  WB health clinic capacity planning tool, NAAH | 0
  WB health clinic capacity planning tool, NA | 20
  Injection flashcard for participants, EH | 2
  Injection flashcard for participants, VH | 7
  Injection flashcard for participants, SH | 2
  Injection flashcard for participants, ALH | 1
  Injection flashcard for participants, NAAH | 0
  Injection flashcard for participants, NA | 11
  Website for participants, EH | 0
  Website for participants, VH | 3
  Website for participants, SH | 3
  Website for participants, ALH | 0
  Website for participants, NAAH | 0
  Website for participants, NA | 17
  What to expect factsheet for participants, EH | 2
  What to expect factsheet for participants, VH | 7
  What to expect factsheet for participants, SH | 6
  What to expect factsheet for participants, ALH | 1
  What to expect factsheet for participants, NAAH | 0
  What to expect factsheet for participants, NA | 7
  Participant handbook, EH | 1
  Participant handbook, VH | 5
  Participant handbook, SH | 5
  Participant handbook, ALH | 2
  Participant handbook, NAAH | 0
  Participant handbook, NA | 10
  FAQs chatbot, EH | 0
  FAQs chatbot, VH | 1
  FAQs chatbot, SH | 0
  FAQs chatbot, ALH | 1
  FAQs chatbot, NAAH | 1
  FAQs chatbot, NA | 20
  Trial guide app, EH | 0
  Trial guide app, VH | 0
  Trial guide app, SH | 0
  Trial guide app, ALH | 0
  Trial guide app, NAAH | 1
  Trial guide app, NA | 22
  Video-what to expect, EH | 4
  Video-what to expect, VH | 7
  Video-what to expect, SH | 3
  Video-what to expect, ALH | 0
  Video-what to expect, NAAH | 0
  Video-what to expect, NA | 9
  Hot and cold packs for participants, EH | 6
  Hot and cold packs for participants, VH | 6
  Hot and cold packs for participants, SH | 6
  Hot and cold packs for participants, ALH | 3
  Hot and cold packs for participants, NAAH | 0
  Hot and cold packs for participants, NA | 2

13. Secondary Outcome: Number of Participants With Change in Barriers to Implementation (BIM) Measure Items Between Baseline and Month 4 Using SSI in Staff Study Participants
Description: BIM is a 23-item survey which assessed barriers (that is, difficulties and challenges) to successful implementation of the CAB LA + RPV LA injection treatment in the study clinic/practices. For each item, providers were asked to rate how much they agreed or disagreed that the issue is a barrier based on their experiences with implementing the CAB + RPV treatment on a five point rating scale (1=completely disagree to 5=completely agree). It is presented as fewer perceived barriers (FPB)=all negative change in scores from Baseline, some perceived barriers (SPB)=change in score of 0 from Baseline, and greater/more perceived barriers (MPB)=all positive change in scores from Baseline.
Time Frame: Baseline and Month 4
Population: All staff study participants population.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 24
Participants
  Interest in the new treatment, FPB | 15
  Interest in the new treatment, SPB | 6
  Interest in the new treatment, MPB | 3
  Incentives for clinical practice change, FPB | 15
  Incentives for clinical practice change, SPB | 3
  Incentives for clinical practice change, MPB | 6
  Ability to keep monthly appointments (apts), FPB | 14
  Ability to keep monthly appointments, SPB | 5
  Ability to keep monthly appointments, MPB | 5
  Failing due to missed doses/injection apts, FPB | 13
  Failing due to missed doses/injection apts, SPB | 9
  Failing due to missed doses/injection apts, MPB | 2
  Lack of familiarity with tools/resources, FPB | 13
  Lack of familiarity with tools/resources, SPB | 8
  Lack of familiarity with tools/resources, MPB | 3
  Transportation for monthly apts, FPB | 12
  Transportation for monthly apts, SPB | 10
  Transportation for monthly apts, MPB | 2
  Injection (Inj)/pain soreness, FPB | 12
  Injection/pain soreness, SPB | 10
  Injection/pain soreness, MPB | 2
  Rescheduling missed injections, FPB | 12
  Rescheduling missed injections, SPB | 9
  Rescheduling missed injections, MPB | 3
  Time for new method implementation CAB+RPV LA, FPB | 12
  Time for new method implementation CAB+RPV LA, SPB | 11
  Time for new method implementation CAB+RPV LA, MPB | 1
  Flagging/awareness of missed injection visits, FPB | 11
  Flagging/awareness of missed injection visits, SPB | 9
  Flagging/awareness of missed injection visits, MPB | 4
  Competing clinic priorities, FPB | 11
  Competing clinic priorities, SPB | 10
  Competing clinic priorities, MPB | 3
  Manage for inj visits with other care need, FPB | 10
  Manage for inj visits with other care need,SPB | 8
  Manage for inj visit with other care need, MPB | 6
  Transition from oral to injection treatment, FPB | 10
  Transition from oral to injection treatment, SPB | 13
  Transition from oral to injection treatment, MPB | 1
  Time to administer the injection, FPB | 10
  Time to administer the injection, SPB | 10
  Time to administer the injection, MPB | 4
  Number of exam rooms for injection, FPB | 9
  Number of exam rooms for injection, SPB | 9
  Number of exam rooms for injection, MPB | 6
  Staff resourcing for clinic flow, FPB | 9
  Staff resourcing for clinic flow, SPB | 8
  Staff resourcing for clinic flow, MPB | 7
  Staff buy-in, FPB | 9
  Staff buy-in, SPB | 13
  Staff buy-in, MPB | 2
  Staff preparation, FPB | 9
  Staff preparation, SPB | 13
  Staff preparation, MPB | 2
  Scheduling of apt reminders, FPB | 8
  Scheduling of apt reminders, SPB | 12
  Scheduling of apt reminders, MPB | 4
  Answering questions between visits, FPB | 7
  Answering questions between visits, SPB | 11
  Answering questions between visits, MPB | 6
  Scheduling of monthly apts, FPB | 7
  Scheduling of monthly apts, SPB | 13
  Scheduling of monthly apts, MPB | 4
  Leadership support, FPB | 6
  Leadership support, SPB | 14
  Leadership support, MPB | 4
  Storage/refrigeration, FPB | 5
  Storage/refrigeration, SPB | 11
  Storage/refrigeration, MPB | 8

14. Secondary Outcome: Percentage of Participants With Change in BIM Measure Items Between Baseline and Month 12 Using SSI in Staff Study Participants
Description: BIM is a 23-item survey which assessed barriers (i.e., difficulties and challenges) to successful implementation of the CAB LA + RPV LA injection treatment in the study clinic/practices. For each item, providers were asked to rate how much they agreed or disagreed that the issue is a barrier based on their experiences with implementing the CAB + RPV treatment on a five point rating scale (1=completely disagree to 5=completely agree). It is presented as fewer perceived barriers (FPB)=all negative change in scores from Baseline, some perceived barriers (SPB)=change in score of 0 from Baseline, and greater/more perceived barriers (MPB)=all positive change in scores from Baseline.
Time Frame: Baseline and Month 12
Population: All staff study participants population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 23
Percentage of participants
  Failing due to missed doses/injection apts, FPB | 78.1
  Failing due to missed doses/injection apts, SPB | 13.0
  Failing due to missed doses/injection apts, MPB | 8.7
  Flagging/awareness of missed injection visits, FPB | 69.5
  Flagging/awareness of missed injection visits, SPB | 26.1
  Flagging/awareness of missed injection visits, MPB | 4.3
  Ability to keep monthly appointments, FPB | 65.2
  Ability to keep monthly appointments, SPB | 34.8
  Ability to keep monthly appointments, MPB | 0.0
  Transportation for monthly apts, FPB | 60.8
  Transportation for monthly apts, SPB | 34.8
  Transportation for monthly apts, MPB | 4.3
  Time for new method implementation CAB+RPV LA, FPB | 60.8
  Time for new method implementation CAB+RPV LA, SPB | 26.1
  Time for new method implementation CAB+RPV LA, MPB | 13.0
  Incentives for clinical practice change, FPB | 60.7
  Incentives for clinical practice change, SPB | 21.7
  Incentives for clinical practice change, MPB | 17.4
  Interest in the new treatment, FPB | 56.5
  Interest in the new treatment, SPB | 26.1
  Interest in the new treatment, MPB | 17.4
  Transition from oral to injection treatment, FPB | 56.5
  Transition from oral to injection treatment, SPB | 39.1
  Transition from oral to injection treatment, MPB | 4.3
  Competing clinic priorities, FPB | 52.1
  Competing clinic priorities, SPB | 43.5
  Competing clinic priorities, MPB | 4.3
  Manage for inj visits with other care need, FPB | 52.1
  Manage for inj visits with other care need,SPB | 43.5
  Manage for inj visit with other care need, MPB | 4.3
  Number of exam rooms for injection, FPB | 52.1
  Number of exam rooms for injection, SPB | 21.7
  Number of exam rooms for injection, MPB | 26.1
  Staff resourcing for clinic flow, FPB | 52.1
  Staff resourcing for clinic flow, SPB | 30.4
  Staff resourcing for clinic flow, MPB | 17.4
  Scheduling of apt reminders, FPB | 52.1
  Scheduling of apt reminders, SPB | 34.8
  Scheduling of apt reminders, MPB | 13.0
  Time to administer the injection, FPB | 47.8
  Time to administer the injection, SPB | 43.5
  Time to administer the injection, MPB | 8.7
  Lack of familiarity with tools/resources, FPB | 47.7
  Lack of familiarity with tools/resources, SPB | 39.1
  Lack of familiarity with tools/resources, MPB | 13.0
  Rescheduling missed injections, FPB | 47.7
  Rescheduling missed injections, SPB | 39.1
  Rescheduling missed injections, MPB | 13.0
  Staff preparation, FPB | 43.4
  Staff preparation, SPB | 47.8
  Staff preparation, MPB | 8.7
  Scheduling of monthly apts, FPB | 43.4
  Scheduling of monthly apts, SPB | 30.4
  Scheduling of monthly apts, MPB | 8.7
  Answering questions between visits, FPB | 39.1
  Answering questions between visits, SPB | 43.5
  Answering questions between visits, MPB | 17.4
  Leadership support, FPB | 39.0
  Leadership support, SPB | 43.5
  Leadership support, MPB | 17.4
  Injection/pain soreness, FPB | 34.8
  Injection/pain soreness, SPB | 56.5
  Injection/pain soreness, MPB | 8.7
  Staff buy-in, FPB | 34.8
  Staff buy-in, SPB | 56.5
  Staff buy-in, MPB | 8.6
  Storage/refrigeration, FPB | 34.8
  Storage/refrigeration, SPB | 43.5
  Storage/refrigeration, MPB | 21.7

15. Secondary Outcome: Number of Participants With HIV Infection Reported Helpfulness of Toolkit Resources at Month 12
Description: The helpfulness of the toolkit resources was identified using a 19-item survey and the helpfulness of the resources were rated on a five point scale where 1=Extremely helpful (EH), 2=Very helpful (VH), 3=Somewhat helpful (SH), 4=A little helpful (ALH) and 5=Not at all helpful (NAAH). Categories for did not receive (DNR) and recevied but did not use (RBDNU) were presented as well. Not Applicable (NA) in the data means participants were not offered the response option. The toolkit resources consisted of information and resources, hot and cold pack, written materials, website for participants, video, verbal information, reminder calls, reminder text messages, reminder app, peer group information session and appointments outside work time. The number of participants with the rating on helpfulness for each toolkit resources is presented.
Time Frame: At Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Participants
  Information and resources, EH | 50
  Information and resources, VH | 40
  Information and resources, SH | 4
  Information and resources, ALH | 2
  Information and resources, NAAH | 0
  Information and resources, DNR | 6
  Information and resources, RBDNU | 0
  Information and resources, Missing | 0
  Hot and cold pack, EH | 18
  Hot and cold pack, VH | 20
  Hot and cold pack, SH | 14
  Hot and cold pack, ALH | 6
  Hot and cold pack, NAAH | 8
  Hot and cold pack, DNR | 9
  Hot and cold pack, RBDNU | 27
  Hot and cold pack, Missing | 0
  Written materials, EH | 37
  Written materials, VH | 37
  Written materials, SH | 11
  Written materials, ALH | 2
  Written materials, NAAH | 0
  Written materials, DNR | 1
  Written materials, RBDNU | 14
  Written materials, Missing | 0
  Website for participants, EH | 25
  Website for participants, VH | 28
  Website for participants, SH | 11
  Website for participants, ALH | 2
  Website for participants, NAAH | 1
  Website for participants, DNR | 4
  Website for participants, RBDNU | 31
  Website for participants, Missing | 0
  Video, EH | 29
  Video, VH | 38
  Video, SH | 13
  Video, ALH | 5
  Video, NAAH | 1
  Video, DNR | 9
  Video, RBDNU | 6
  Video, Missing | 1
  Verbal information, EH | 69
  Verbal information, VH | 31
  Verbal information, SH | 2
  Verbal information, ALH | 0
  Verbal information, NAAH | 0
  Verbal information, DNR | 0
  Verbal information, RBDNU | 0
  Verbal information, Missing | 0
  Reminder calls, EH | 67
  Reminder calls, VH | 24
  Reminder calls, SH | 5
  Reminder calls, ALH | 1
  Reminder calls, NAAH | 1
  Reminder calls, DNR | 4
  Reminder calls, RBDNU | 0
  Reminder calls, Missing | 0
  Reminder text messages, EH | 63
  Reminder text messages, VH | 19
  Reminder text messages, SH | 4
  Reminder text messages, ALH | 1
  Reminder text messages, NAAH | 0
  Reminder text messages, DNR | 15
  Reminder text messages, RBDNU | 0
  Reminder text messages, Missing | 0
  Reminder app, EH | 26
  Reminder app, VH | 14
  Reminder app, SH | 3
  Reminder app, ALH | 0
  Reminder app, NAAH | 0
  Reminder app, DNR | 28
  Reminder app, RBDNU | 31
  Reminder app, Missing | 0
  Peer group informational (info) session, EH | 24
  Peer group info session, VH | 27
  Peer group info session, SH | 25
  Peer group info session, ALH | 6
  Peer group info session, NAAH | 20
  Peer group info session, DNR | NA — Participants were not offered the response option.
  Peer group info session, RBDNU | NA — Participants were not offered the response option.
  Peer group info session, Missing | 0
  Apts outside work time, EH | 63
  Apts outside work time, VH | 22
  Apts outside work time, SH | 13
  Apts outside work time, ALH | 1
  Apts outside work time, NAAH | 3
  Apts outside work time, DNR | NA — Participants were not offered the response option.
  Apts outside work time, RBDNU | NA — Participants were not offered the response option.
  Apts outside work time, Missing | 0

16. Secondary Outcome: Number of Participants With HIV Reporting Barriers to CAB LA + RPV LA Injection Treatment at Month 12
Description: Participants were asked to report any factors that were interfering with their ability to get the monthly CAB LA + RPV LA injection treatment. Number of participants along with the reasons for interference in ability to get CAB LA + RPV LA is presented.
Time Frame: At Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Participants
  Pain or soreness from the injection | 15
  Scheduling upcoming injection visits | 2
  Rescheduling missed injection visits | 1
  Forgetting appointment for the injection visits | 2
  Frequency of required visits to clinic for inj | 6
  Missing work too frequently for the injection | 7
  Transportation to clinic/practice for inj visit | 3
  Ease of parking at clinic/practice for inj visit | 4
  Limited clinic/practice hours for inj visits | 3
  Less privacy for inj visits than daily HIV medicine | 1
  Nothing is interfering with getting this treatment | 75

17. Secondary Outcome: Number of Barriers Assessed Among Clinics Using Short-term Facilitation
Description: The barriers were analyzed using semi-structured interviews from the validated consolidated framework for implementation research (CFIR) across 7 calls. An implementation science approach was used to understand the barriers for participants with HIV for delivering CAB + RPV LA within an interventional clinical trial where the CAB + RPV LA regimen was delivered to HIV infected, virologically-suppressed participants.
Time Frame: Up to 6 months
Population: Safety population
Measure: Number; unit: Barriers
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Barriers
  Facilitation call 1 | 5
  Facilitation call 2 | 3
  Facilitation call 3 | 7
  Facilitation call 4 | 6
  Facilitation call 5 | 4
  Facilitation call 6 | 7
  Facilitation call 7 | 3

18. Secondary Outcome: Number of Facilitators Assessed Among Clinics Using Short-term Facilitation
Description: The facilitators were analyzed using semi-structured interviews from the validated CFIR across 7 calls. An implementation science approach was used to understand the facilitators for participants with HIV for delivering CAB + RPV LA within an interventional clinical trial where the CAB + RPV LA regimen was delivered to HIV infected, virologically-suppressed participants.
Time Frame: Up to 6 months
Population: Safety population
Measure: Number; unit: Facilitators
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Facilitators
  Facilitation call 1 | 7
  Facilitation call 2 | 3
  Facilitation call 3 | 3
  Facilitation call 4 | 5
  Facilitation call 5 | 9
  Facilitation call 6 | 9
  Facilitation call 7 | 8

19. Secondary Outcome: Number of Best Practices Assessed Among Clinics Using Short-term Facilitation
Description: The best practices were analyzed using short-term facilitation calls. An implementation science approach was used to understand the best practices for participants with HIV for delivering CAB + RPV LA within an interventional clinical trial where the CAB + RPV LA regimen was delivered to HIV infected, virologically-suppressed participants.
Time Frame: Up to 6 months
Population: Safety population
Measure: Number; unit: Best practices
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Best practices
  Facilitation call 1 | 5
  Facilitation call 2 | 2
  Facilitation call 3 | 2
  Facilitation call 4 | 5
  Facilitation call 5 | 6
  Facilitation call 6 | 6
  Facilitation call 7 | 8

20. Secondary Outcome: Number of Staff Study Participants Using Support Materials/Toolkit at Month 4
Description: Number of staff study participants using support materials/toolkit at Month 4 was assessed by variables: Not used, Used similar resource, used the support materials/toolkit. The support materials/toolkit consisted of website for clinical staff, video on giving CAB + RPV LA, how to use new packaging card, study factsheet for healthcare providers, consultation aid, reminder e-application, reminder SMS/text, face-to-face training by healthcare staff, facilitation group calls, web-based (WB) treatment planner, WB health clinic capacity planning tool, injection flashcards, website for participants, what to expect factsheet for participants, handbook, FAQ chatbot, trial guide app, video-what to expect and hot and cold packs.
Time Frame: At Month 4
Population: All Staff study participants population
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 24
Participants
  Website for clinical staff, not used | 9
  Website for clinical staff, used similar | 1
  Website for clinical staff, used | 14
  Video on giving CAB + RPV LA injection, not used | 8
  Video on giving CAB + RPV LA injection, used similar | 1
  Video on giving CAB + RPV LA injection, used | 15
  How to use new packaging card, not used | 11
  How to use new packaging card, used similar | 0
  How to use new packaging card, used | 13
  Study factsheet for HCP, not used | 8
  Study factsheet for HCP, used similar | 1
  Study factsheet for HCP, used | 15
  Consultation aid, not used | 12
  Consultation aid, used similar | 1
  Consultation aid, used | 11
  Reminder, e-app, not used | 16
  Reminder e-app, used similar | 2
  Reminder e-app, used | 6
  Reminder SMS/text, not used | 15
  Reminder SMS/text, used similar | 4
  Reminder SMS/text, used | 5
  F2F training, not used | 8
  F2F training, used similar | 1
  F2F training, used | 15
  Facilitation group calls, not used | 4
  Facilitation group calls, used similar | 1
  Facilitation group calls, used | 19
  WB treatment planner, not used | 12
  WB treatment planner, used similar | 0
  WB treatment planner, used | 12
  WB health clinic capacity planning tool, not used | 20
  WB health clinic planning tool, used similar | 2
  WB health clinic capacity planning tool, used | 2
  Injection flashcard, not used | 10
  Injection flashcard, used similar | 2
  Injection flashcard, used | 12
  Website for participants, not used | 14
  Website for participants, used similar | 1
  Website for participants, used | 9
  What to expect factsheet, not used | 8
  What to expect factsheet, used similar | 1
  What to expect factsheet, used | 15
  Participant handbook, not used | 12
  Participant handbook, used similar | 0
  Participant handbook, used | 12
  FAQ chatbot, not used | 18
  FAQ chatbot, used similar | 0
  FAQ chatbot, used | 6
  Trial guide app, not used | 19
  Trail guide app, used similar | 0
  Trial guide app, used | 5
  Video-what to expect, not used | 8
  Video-what to expect, used similar | 0
  Video-what to expect, used | 16
  Hot and cold pack, not used | 6
  Hot and cold pack, used similar | 0
  Hot and cold pack, used | 18

21. Secondary Outcome: Number of Staff Study Participants Using Support Materials/Toolkit at Month 12
Description: Number of staff study participants using support materials/toolkit at Month 12 was assessed by variables: Not used, Used similar resource, used the support materials/toolkit. The support materials/toolkit consisted of website for clinical staff, video on giving CAB + RPV LA, how to use new packaging card, study factsheet for healthcare providers, consultation aid, reminder e-application, reminder SMS/text, face-to-face training by healthcare staff, facilitation group calls, web-based (WB) treatment planner, WB health clinic capacity planning tool, injection flashcards, website for participants, what to expect factsheet for participants, handbook, FAQ chatbot, trial guide app, video-what to expect and hot and cold packs.
Time Frame: At Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 23
Participants
  Website for clinical staff, not used | 13
  Website for clinical staff, used similar | 0
  Website for clinical staff, used | 10
  Video on giving CAB + RPV LA injection, not used | 6
  Video on giving CAB + RPV LA injection, used similar | 0
  Video on giving CAB + RPV LA injection, used | 17
  How to use new packaging card, not used | 14
  How to use new packaging card, used similar | 0
  How to use new packaging card, used | 9
  Study factsheet for HCP, not used | 10
  Study factsheet for HCP, used similar | 1
  Study factsheet for HCP, used | 12
  Consultation aid, not used | 14
  Consultation aid, used similar | 0
  Consultation aid, used | 9
  Reminder, e-app, not used | 15
  Reminder e-app, used similar | 6
  Reminder e-app, used | 2
  Reminder SMS/text, not used | 8
  Reminder SMS/text, used similar | 10
  Reminder SMS/text, used | 5
  F2F training, not used | 3
  F2F training, used similar | 1
  F2F training, used | 19
  Facilitation group calls, not used | 6
  Facilitation group calls, used similar | 1
  Facilitation group calls, used | 16
  WB treatment planner, not used | 11
  WB treatment planner, used similar | 2
  WB treatment planner, used | 10
  WB health clinic capacity planning tool, not used | 16
  WB health clinic planning tool, used similar | 4
  WB health clinic capacity planning tool, used | 3
  Injection flashcard, not used | 9
  Injection flashcard, used similar | 2
  Injection flashcard, used | 12
  Website for participants, not used | 15
  Website for participants, used similar | 2
  Website for participants, used | 6
  What to expect factsheet, not used | 5
  What to expect factsheet, used similar | 2
  What to expect factsheet, used | 16
  Participant handbook, not used | 8
  Participant handbook, used similar | 2
  Participant handbook, used | 13
  FAQ chatbot, not used | 18
  FAQ chatbot, used similar | 2
  FAQ chatbot, used | 3
  Trial guide app, not used | 20
  Trail guide app, used similar | 2
  Trial guide app, used | 1
  Video-what to expect, not used | 8
  Video-what to expect, used similar | 1
  Video-what to expect, used | 14
  Hot and cold pack, not used | 2
  Hot and cold pack, used similar | 0
  Hot and cold pack, used | 21

22. Secondary Outcome: Percentage of Participants With HIV Reporting Helpfulness of the Use of Support Materials/Toolkit at Month 4
Description: Participants with HIV infection were asked about their utilization of each element of the support materials/toolkit and were asked to categorize it as Extremely helpful (EH) Very helpful (VH), Somewhat helpful (SH), A little helpful (ALH), Not at all helpful (NAAH), did not receive (DNR), Received but did not use (RBDNU) and missing. Not Applicable (NA) in the data means participants were not offered the response option. The support materials/toolkit consisted of information and resources, hot and cold pack, written materials, website for participants, video, verbal information, reminder calls, reminder text messages, reminder app, peer group information session and appointments outside work time. Percentage of participants with the rating on helpfulness for each toolkit resources is presented.
Time Frame: At Month 4
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 105
Percentage of participants
  Information and resources, EH | 49.5
  Information and resources, VH | 38.1
  Information and resources, SH | 6.7
  Information and resources, ALH | 1.9
  Information and resources, NAAH | 0.0
  Information and resources, DNR | 3.8
  Information and resources, RBDNU | 0.0
  Information and resources, Missing | 0.0
  Hot and cold pack, EH | 19.0
  Hot and cold pack, VH | 8.6
  Hot and cold pack, SH | 21.9
  Hot and cold pack, ALH | 8.6
  Hot and cold pack, NAAH | 2.9
  Hot and cold pack, DNR | 14.3
  Hot and cold pack, RBDNU | 23.8
  Hot and cold pack, Missing | 1.0
  Written materials, EH | 38.1
  Written materials, VH | 35.2
  Written materials, SH | 12.4
  Written materials, ALH | 1.9
  Written materials, NAAH | 1.0
  Written materials, DNR | 1.9
  Written materials, RBDNU | 9.5
  Written materials, Missing | 0.0
  Website, EH | 21.0
  Website, VH | 28.6
  Website, SH | 5.7
  Website, ALH | 1.9
  Website, NAAH | 1.9
  Website, DNR | 6.7
  Website, RBDNU | 34.3
  Website, Missing | 0.0
  Video, EH | 28.6
  Video, VH | 41.0
  Video, SH | 12.4
  Video, ALH | 4.8
  Video, NAAH | 1.9
  Video, DNR | 8.6
  Video, RBDNU | 2.9
  Video, Missing | 0.0
  Verbal information, EH | 62.9
  Verbal information, VH | 32.4
  Verbal information, SH | 3.8
  Verbal information, ALH | 0.0
  Verbal information, NAAH | 0.0
  Verbal information, DNR | 0.0
  Verbal information, RBDNU | 0.0
  Verbal information, Missing | 1.0
  Reminder calls, EH | 61.0
  Reminder calls, VH | 23.8
  Reminder calls, SH | 4.8
  Reminder calls, ALH | 4.8
  Reminder calls, NAAH | 0.0
  Reminder calls, DNR | 4.8
  Reminder calls, RBDNU | 0.0
  Reminder calls, Missing | 1.0
  Reminder text messages, EH | 56.2
  Reminder text messages, VH | 19.0
  Reminder text messages, SH | 4.8
  Reminder text messages, ALH | 1.0
  Reminder text messages, NAAH | 0.0
  Reminder text messages, DNR | 18.1
  Reminder text messages, RBDNU | 0.0
  Reminder text messages, Missing | 1.0
  Reminder app, EH | 23.8
  Reminder app, VH | 16.2
  Reminder app, SH | 2.9
  Reminder app, ALH | 1.9
  Reminder app, NAAH | 0.0
  Reminder app, DNR | 26.7
  Reminder app, RBDNU | 28.6
  Reminder app, Missing | 0.0
  Peer group informational (info) session, EH | 22.9
  Peer group info session, VH | 20.0
  Peer group info session, SH | 33.3
  Peer group info session, ALH | 8.6
  Peer group info session, NAAH | 14.3
  Peer group info session, DNR | NA — Participants were not offered the response option.
  Peer group info session, RBDNU | NA — Participants were not offered the response option.
  Peer group info session, Missing | 1.0
  Apts outside work time, EH | 57.1
  Apts outside work time, VH | 26.7
  Apts outside work time, SH | 6.7
  Apts outside work time, ALH | 4.8
  Apts outside work time, NAAH | 4.8
  Apts outside work time, DNR | NA — Participants were not offered the response option.
  Apts outside work time, RBDNU | NA — Participants were not offered the response option.
  Apts outside work time, Missing | 0.0

23. Secondary Outcome: Number of Participants Receiving Injections Within Target Window at Month 4
Description: Number of participants receiving injections within target window at Month 4 is presented. The target window is +/- 7 days from the target injection visit date.
Time Frame: At Month 4
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 105
Participants | 100

24. Secondary Outcome: Number of Participants Receiving Injections Within Target Window at Month 12
Description: Number of participants receiving injections within target window at Month 12 is presented. The target window is +/- 7 days from the target injection visit date.
Time Frame: At Month 12
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Participants | 96

25. Secondary Outcome: Implementation Sustainability Assessed in Staff Study Participants Using Program Sustainability Assessment Tool (PSAT) Scores
Description: Implementation sustainability in staff study participants was assessed using PSAT tool that evaluated capability of clinics to maintain processes developed to administer CAB+RPV injection in routine clinical settings after study conclusion.It consisted of 6 domains(1.Environmental support,2.Organizational capacity,3.Program evaluation,4.Program adaptation,5.Communications and 6.Strategic planning).Each domain consisted of 5 items,each assessed using 7-point numerical rating scale:1=to not extent at all,7=to a very great extent and an eighth not applicable/not able to answer response(NA).Score ranges for total domain scores are 5 to 35 for each of 6 domains(5 items in each domain on 1 to 7 scale).Numeric response to each item within specific domain is summed to produce a total domain score then mean domain score is calculated(excluding any NA responses).Higher scores indicate better outcome(higher endorsement/more positive impressions by staff-study with sustainability survey concepts)
Time Frame: At Month 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants
Number analyzed (Participants) | 23
Scores on a scale
  Environmental support | 5.82 (0.20)
  Organizational capacity | 5.74 (0.28)
  Program evaluation | 5.83 (0.49)
  Program adaptation | 5.98 (0.15)
  Communications | 6.09 (0.06)
  Strategic planning | 5.50 (0.34)

26. Secondary Outcome: HIV Treatment Satisfaction Questionnaire Status Version (HIV-TSQs) Scores at Month 1
Description: Participant satisfaction was measured using the validated HIV Treatment Satisfaction Questionnaire (HIV-TSQ), status version (HIV-TSQs), which measured satisfaction with the treatment used in the previous few weeks. HIVTSQs total treatment satisfaction score was computed with 1-11 items. Each item was scored from 0 (least satisfied) to 6 (most satisfied). Items 1-11 were summed to produce score with possible range of 0 to 66. Higher the score, greater improvement in satisfaction with treatment; lower score, greater the deterioration in satisfaction with treatment.
Time Frame: At Month 1
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 109
Scores on a scale | 60.7 (6.3)

27. Secondary Outcome: HIV-TSQs Scores at Month 4
Description: as for outcome 26
Time Frame: At Month 4
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 105
Scores on a scale | 62.12 (5.79)

28. Secondary Outcome: HIV-TSQs Scores at Month 12
Description: as for outcome 26
Time Frame: At Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Scores on a scale | 63.30 (3.81)

29. Secondary Outcome: Number of Participants With Reported Acceptability of the Amount of Time Spent in the Clinic for Each Injection Visit
Description: The results for participant reported acceptability of the amount of time spent in the clinic for each injection visit is presented. Participants were asked to rate the acceptability of the amount of time spent in the clinic for each injection visit as extremely acceptable, very acceptable, somewhat acceptable, a little acceptable and not at all acceptable.
Time Frame: At Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Participants
  Extremely acceptable | 62
  Very acceptable | 33
  Somewhat acceptable | 7
  A little acceptable | 0
  Not at all acceptable | 0

30. Secondary Outcome: Number of Participants With the Reported Time Spent in Clinic/Practice for Each Injection Visit
Description: Number of participants with the reported time spent in clinic/practice for each injection visit is presented.
Time Frame: At Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Participants
  1-15 minutes | 14
  16-30 minutes | 51
  31-45 minutes | 23
  46-60 minutes | 12
  More than 60 minutes | 1

31. Secondary Outcome: Number of Participants With Extent of Knowledge About the CAB + RPV LA Treatment
Description: Participants were asked to rate how knowledgeable they feel about the CAB LA + RPV LA treatment as extremely knowledgeable, very knowledgeable, somewhat knowledgeable, a little knowledgeable and not at all knowledgeable.
Time Frame: At Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 102
Participants
  Extremely knowledgeable | 34
  Very knowledgeable | 40
  Somewhat knowledgeable | 25
  A little knowledgeable | 2
  Not at all knowledgeable | 1

32. Secondary Outcome: Length of Participant Visit
Description: Length of visit was calculated by subtracting the arrival time (Lead time [actual start time of appointment - arrival time] + process time [actual end time of appointment - actual start time of appointment]) from actual end time of appointment.
Time Frame: At Months 1, 5 and 11
Population: Safety population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Minutes
  At Month 1, n=109: number analyzed (Participants) | 109
  At Month 1, n=109 | 63.4 (29.51)
  At Month 5, n=104: number analyzed (Participants) | 104
  At Month 5, n=104 | 38.7 (19.91)
  At Month 11, n=100: number analyzed (Participants) | 100
  At Month 11, n=100 | 36.3 (16.85)

33. Secondary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) Less Than (<)50 Copies/Milliliter (c/mL) by Modified Food and Drug Administration (FDA) Snapshot Algorithm
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with plasma HIV-1 RNA <50 c/mL (virologic success) was evaluated using the modified Food and Drug Administration (FDA) snapshot algorithm with Coronavirus Disease 2019 (COVID-19) related missing value imputed using the last observation carried forward (LOCF) approach.
Time Frame: Month 1, Month 2, Month 4, Month 6, Month 8, Month 10 and Month 12
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Percentage of participants
  Month 1 | 93.9
  Month 2 | 94.8
  Month 4 | 91.3
  Month 6 | 90.4
  Month 8 | 88.7
  Month 10 | 87.8
  Month 12 | 88.7

34. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL - Observed Case
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. The percentage value presented has been rounded off.
Time Frame: Months 1, Month 2, Month 4, Month 6, Month 8, Month 10, Month 12, Month 13, Month 15, Month 16, Month 18, Month 19, Month 21, Month 22, Month 24, Month 25, Month 27, Month 28 and Month 30
Population: as for outcome 32
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Percentage of participants
  Month 1; n=112: number analyzed (Participants) | 112
  Month 1; n=112 | 96
  Month 2; n=109: number analyzed (Participants) | 109
  Month 2; n=109 | 100
  Month 4; n=107: number analyzed (Participants) | 107
  Month 4; n=107 | 98
  Month 6; n=103: number analyzed (Participants) | 103
  Month 6; n=103 | 100
  Month 8; n=94: number analyzed (Participants) | 94
  Month 8; n=94 | 100
  Month 10; n=100: number analyzed (Participants) | 100
  Month 10; n=100 | 99
  Month 12, n=101: number analyzed (Participants) | 101
  Month 12, n=101 | 100
  Month 13; n=101: number analyzed (Participants) | 101
  Month 13; n=101 | 100
  Month 15; n=99: number analyzed (Participants) | 99
  Month 15; n=99 | 100
  Month 16; n=94: number analyzed (Participants) | 94
  Month 16; n=94 | 99
  Month 18; n=95: number analyzed (Participants) | 95
  Month 18; n=95 | 100
  Month 19; n=89: number analyzed (Participants) | 89
  Month 19; n=89 | 100
  Month 21; n=75: number analyzed (Participants) | 75
  Month 21; n=75 | 100
  Month 22; n=61: number analyzed (Participants) | 61
  Month 22; n=61 | 100
  Month 24; n=35: number analyzed (Participants) | 35
  Month 24; n=35 | 100
  Month 25; n=17: number analyzed (Participants) | 17
  Month 25; n=17 | 100
  Month 27; n=8: number analyzed (Participants) | 8
  Month 27; n=8 | 100
  Month 28; n=7: number analyzed (Participants) | 7
  Month 28; n=7 | 100
  Month 30; n=1: number analyzed (Participants) | 1
  Month 30; n=1 | 100

35. Secondary Outcome: Percentage of Participants With Confirmed Virologic Failure (CVF)
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. The CVF is defined as rebound as indicated by two consecutive plasma HIV-1 RNA levels greater than or equal to (>=)200 copies/mL after prior suppression to <200 copies/mL.
Time Frame: Up to 30 months
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Percentage of participants | 0

36. Secondary Outcome: Number of Participants With Treatment Emergent Genotypic Resistance to CAB and RPV
Description: Plasma samples were collected for drug resistance testing. Number of participants who met CVF criteria (two consecutive plasma HIV-1 RNA levels >=200 copies/mL after prior suppression to <200 copies/mL) with emergent genotypic resistance is summarized.
Time Frame: Up to 30 months
Population: Safety population. Only participants with CVF were included in the analysis
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 0

37. Secondary Outcome: Number of Participants With Treatment Emergent Phenotypic Resistance to CAB and RPV
Description: Plasma samples were collected for drug resistance testing. Number of participants who met CVF criteria (two consecutive plasma HIV-1 RNA levels >=200 copies/mL after prior suppression to <200 copies/mL) with emergent phenotypic resistance is summarized.
Time Frame: Up to 30 months
Population: Safety population. Only participants with CVF were included in the analysis
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 0

38. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Common (>=5 Percent [%]) Non-serious Adverse Events (Non-SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose may result in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function. Number of participants with any SAE and common (>=5%) non-SAEs are presented. Adverse events which were not serious have been considered as non-serious adverse events.
Time Frame: Up to 30 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants
  Common (>=5%) non-SAEs | 101
  SAEs | 9

39. Secondary Outcome: Percentage of Participants Who Discontinue Treatment or Withdraw From Study Due to AEs Over Time
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Percentage of participants with adverse events leading to study treatment or study withdrawal has been presented. The percentage value presented has been rounded off.
Time Frame: Up to 30 months
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Percentage of participants | 7

40. Secondary Outcome: Number of Participants With Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of following hematology parameters: leukocytes, neutrophils and platelets. The parameters were graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scale from Grade 1 to 4, where Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). Higher the grade, more severe the symptoms.
Time Frame: Up to Month 12
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants
  Leukocytes, increase from Grade 1 to 4 | 5
  Leukocytes, increase from Grade 2 to 4 | 2
  Leukocytes, increase from Grade 3 to 4 | 1
  Neutrophils, increase from Grade 1 to 4 | 8
  Neutrophils, increase from Grade 2 to 4 | 3
  Neutrophils, increase from Grade 3 to 4 | 1
  Platelets, increase from Grade 1 to 4 | 1
  Platelets, increase from Grade 2 to 4 | 0
  Platelets, increase from Grade 3 to 4 | 0

41. Secondary Outcome: Number of Participants With Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline Through End of Study
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin, leukocytes, neutrophils and platelets. The parameters were graded according to the DAIDS toxicity scale from Grade 1 to 4, where Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). Higher the grade, more severe the symptoms.
Time Frame: Up to 30 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants
  Hemoglobin, increase from Grades 1 to 4 | 1
  Hemoglobin, increase from Grades 2 to 4 | 0
  Hemoglobin, increase from Grades 3 to 4 | 0
  Leukocytes, increase from Grade 1 to 4 | 6
  Leukocytes, increase from Grade 2 to 4 | 2
  Leukocytes, increase from Grade 3 to 4 | 1
  Neutrophils, increase from Grade 1 to 4 | 9
  Neutrophils, increase from Grade 2 to 4 | 4
  Neutrophils, increase from Grade 3 to 4 | 2
  Platelets, increase from Grade 1 to 4 | 2
  Platelets, increase from Grade 2 to 4 | 0
  Platelets, increase from Grade 3 to 4 | 0

42. Secondary Outcome: Number of Participants With Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected up to the Month 12 visit for the analysis of clinical chemistry parameters: alanine aminotransferase (ALT), alkaline phosphate (ALP), aspartate aminotransferase (AST), bilirubin, carbon dioxide (CO2), creatine kinase (CK), creatinine, direct bilirubin, glucose, lipase, phosphate, potassium and sodium. Any abnormality in clinical chemistry parameters were evaluated according to the DAIDS toxicity scale From Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). Higher the grade, more severe the symptoms.
Time Frame: Up to Month 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants
  ALT, increase from Grade 1 to 4 | 15
  ALT, increase from Grade 2 to 4 | 3
  ALT, increase from Grade 3 to 4 | 0
  ALP, increase from Grade 1 to 4 | 3
  ALP, increase from Grade 2 to 4 | 0
  ALP, increase from Grade 3 to 4 | 0
  AST, increase from Grade 1 to 4 | 8
  AST, increase from Grade 2 to 4 | 4
  AST, increase from Grade 3 to 4 | 0
  Bilirubin, increase from Grade 1 to 4 | 4
  Bilirubin, increase from Grade 2 to 4 | 1
  Bilirubin, increase from Grade 3 to 4 | 0
  CO2, increase from Grade 1 to 4 | 16
  CO2, increase from Grade 2 to 4 | 0
  CO2, increase from Grade 3 to 4 | 0
  CK, increase from Grade 1 to 4 | 11
  CK, increase from Grade 2 to 4 | 4
  CK, increase from Grade 3 to 4 | 1
  Creatinine, increase from Grade 1 to 4 | 2
  Creatinine, increase from Grade 2 to 4 | 1
  Creatinine, increase from Grade 3 to 4 | 0
  Direct bilirubin, increase from Grade 1 to 4 | 1
  Direct bilirubin, increase from Grade 2 to 4 | 1
  Direct bilirubin, increase from Grade 3 to 4 | 1
  Glucose, increase from Grade 1 to 4 | 18
  Glucose, increase from Grade 2 to 4 | 8
  Glucose, increase from Grade 3 to 4 | 0
  Lipase, increase from Grade 1 to 4 | 17
  Lipase, increase from Grade 2 to 4 | 11
  Lipase, increase from Grade 3 to 4 | 0
  Phosphate, increase from Grade 1 to 4 | 16
  Phosphate, increase from Grade 2 to 4 | 4
  Phosphate, increase from Grade 3 to 4 | 0
  Potassium, increase from Grade 1 to 4 | 4
  Potassium, increase from Grade 2 to 4 | 0
  Potassium, increase from Grade 3 to 4 | 0
  Sodium, increase from Grade 1 to 4 | 6
  Sodium, increase from Grade 2 to 4 | 0
  Sodium, increase from Grade 3 to 4 | 0

43. Secondary Outcome: Number of Participants With Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline Through End of Study
Description: Blood samples were collected for the analysis of clinical chemistry parameters: ALT, ALP, AST, bilirubin, CO2, CK, creatinine, direct bilirubin, Glomerular filtration rate (GFR) from Creatinine (Creat) Adjusted (Adj) using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), GFR From Creat Adj for body surface area (BSA), glucose, lipase, phosphate, potassium and sodium. Any abnormality in clinical chemistry parameters were evaluated according to the DAIDS toxicity scale From Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). Higher the grade, more severe the symptoms.
Time Frame: Up to 30 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants
  ALT, increase from Grade 1 to 4 | 24
  ALT, increase from Grade 2 to 4 | 6
  ALT, increase from Grade 3 to 4 | 0
  ALP, increase from Grade 1 to 4 | 3
  ALP, increase from Grade 2 to 4 | 0
  ALP, increase from Grade 3 to 4 | 0
  AST, increase from Grade 1 to 4 | 13
  AST, increase from Grade 2 to 4 | 5
  AST, increase from Grade 3 to 4 | 1
  Bilirubin, increase from Grade 1 to 4 | 6
  Bilirubin, increase from Grade 2 to 4 | 1
  Bilirubin, increase from Grade 3 to 4 | 0
  CO2, increase from Grade 1 to 4 | 18
  CO2, increase from Grade 2 to 4 | 0
  CO2, increase from Grade 3 to 4 | 0
  CK, increase from Grade 1 to 4 | 18
  CK, increase from Grade 2 to 4 | 9
  CK, increase from Grade 3 to 4 | 4
  Creatinine, increase from Grade 1 to 4 | 5
  Creatinine, increase from Grade 2 to 4 | 1
  Creatinine, increase from Grade 3 to 4 | 0
  Direct bilirubin, increase from Grade 1 to 4 | 1
  Direct bilirubin, increase from Grade 2 to 4 | 1
  Direct bilirubin, increase from Grade 3 to 4 | 1
  GFR From Creat Adj Using CKD-EPI increase from Grade 1 to 4 | 27
  GFR From Creat Adj Using CKD-EPI increase from Grade 2 to 4 | 27
  GFR From Creat Adj Using CKD-EPI increase from Grade 3 to 4 | 6
  GFR From Creat Adj for BSA increase from Grade 1 to 4 | 27
  GFR From Creat Adj for BSA increase from Grade 2 to 4 | 27
  GFR From Creat Adj for BSA increase from Grade 3 to 4 | 6
  Glucose, increase from Grade 1 to 4 | 26
  Glucose, increase from Grade 2 to 4 | 16
  Glucose, increase from Grade 3 to 4 | 2
  Lipase, increase from Grade 1 to 4 | 23
  Lipase, increase from Grade 2 to 4 | 16
  Lipase, increase from Grade 3 to 4 | 0
  Phosphate, increase from Grade 1 to 4 | 22
  Phosphate, increase from Grade 2 to 4 | 6
  Phosphate, increase from Grade 3 to 4 | 0
  Potassium, increase from Grade 1 to 4 | 4
  Potassium, increase from Grade 2 to 4 | 0
  Potassium, increase from Grade 3 to 4 | 0
  Sodium, increase from Grade 1 to 4 | 7
  Sodium, increase from Grade 2 to 4 | 0
  Sodium, increase from Grade 3 to 4 | 0

44. Secondary Outcome: Number of Participants With Urinalysis Result of Potential Clinical Importance
Description: Urine samples were collected to analyze the urine parameters: Protein, occult blood or glucose. Potential clinical importance is defined as an increase in protein (dipstick) or occult blood (dipstick) post-Baseline relative to Baseline. Number of participants with results of potential clinical importance in any of the urine parameters is presented.
Time Frame: Up to Month 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants | 8

45. Secondary Outcome: Number of Participants With Urinalysis Result of Potential Clinical Importance Through End of Study
Description: as for outcome 44
Time Frame: Up to 30 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants | 1

46. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) Over Time
Description: Local tolerability was measured by injection site reaction (ISR), for example; bruise at the site of injection and/or itching, pain, blistering or skin damage. ISRs were assigned to the most recent planned injection visit prior to/on the onset date of the ISR. Number of participants with ISRs by each assigned injection visit is presented.
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants
  Month 1 | 109
  Month 2 | 108
  Month 3 | 106
  Month 4 | 105
  Month 5 | 104
  Month 6 | 103
  Month 7 | 103
  Month 8 | 102
  Month 9 | 100
  Month 10 | 100
  Month 11 | 100
  Month 12 | 101

47. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) Over Time From Month 13 to Month 30
Description: as for outcome 46
Time Frame: Months 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29 and 30
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Participants
  Month 13 | 99
  Month 14 | 99
  Month 15 | 98
  Month 16 | 96
  Month 17 | 95
  Month 18 | 97
  Month 19 | 95
  Month 20 | 86
  Month 21 | 75
  Month 22 | 65
  Month 23 | 49
  Month 24 | 35
  Month 25 | 19
  Month 26 | 11
  Month 27 | 8
  Month 28 | 7
  Month 29 | 4
  Month 30 | 1

48. Secondary Outcome: Change From Baseline in Hematology Parameters: Platelet Count, White Blood Cell (WBC) Count, Basophil Count, Eosinophil Count, Lymphocyte Count, Monocyte Count and Neutrophil Count
Description: Blood samples were collected to analyze the hematology parameters: Platelet count, WBC count, Basophil count, Eosinophil count, Lymphocyte count, Monocyte count and Neutrophil count. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
10^9 cells per Liter
  Platelet count, n=100: number analyzed (Participants) | 100
  Platelet count, n=100 | -0.66 (33.512)
  WBC count, n=101: number analyzed (Participants) | 101
  WBC count, n=101 | 0.27 (1.412)
  Basophil count, n=101: number analyzed (Participants) | 101
  Basophil count, n=101 | 0.006 (0.0232)
  Eosinophil count, n=101: number analyzed (Participants) | 101
  Eosinophil count, n=101 | 0.018 (0.1632)
  Lymphocyte count, n=101: number analyzed (Participants) | 101
  Lymphocyte count, n=101 | -0.0005 (0.49237)
  Monocyte count, n=101: number analyzed (Participants) | 101
  Monocyte count, n=101 | 0.029 (0.1434)
  Neutrophil count, n=101: number analyzed (Participants) | 101
  Neutrophil count, n=101 | 0.214 (1.1746)

49. Secondary Outcome: Change From Baseline in Hematology Parameter: Red Blood Cell (RBC) Count
Description: Blood samples were collected to analyze the hematology parameter: RBC count. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
10^12 cells per liter | 0.18 (0.260)

50. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Grams per liter | -1.11 (7.221)

51. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit (fraction of 1). Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Percentage of red blood cells in blood | -0.0022 (0.02554)

52. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume (MCV)
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes MCV. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Femtoliter | -3.90 (2.961)

53. Secondary Outcome: Change From Baseline in Hematology Parameters: Platelet Count, White Blood Cell (WBC) Count, Basophil Count, Eosinophil Count, Lymphocyte Count , Monocyte Count and Neutrophil Count From Month 15 to Month 30
Description: as for outcome 48
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
10^9 cells per Liter
  Platelet count, Month 15, n=98: number analyzed (Participants) | 98
  Platelet count, Month 15, n=98 | 5.47 (41.191)
  Platelet count, Month 18, n=96: number analyzed (Participants) | 96
  Platelet count, Month 18, n=96 | 9.59 (57.934)
  Platelet count, Month 21, n=75: number analyzed (Participants) | 75
  Platelet count, Month 21, n=75 | 8.07 (34.613)
  Platelet count, Month 24, n=35: number analyzed (Participants) | 35
  Platelet count, Month 24, n=35 | 14.51 (24.923)
  Platelet count, Month 27, n=8: number analyzed (Participants) | 8
  Platelet count, Month 27, n=8 | 31.13 (48.265)
  Platelet count, Month 30, n=1: number analyzed (Participants) | 1
  Platelet count, Month 30, n=1 | 73.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  WBC count, Month 15, n=99: number analyzed (Participants) | 99
  WBC count, Month 15, n=99 | 0.66 (1.648)
  WBC count, Month 18, n=97: number analyzed (Participants) | 97
  WBC count, Month 18, n=97 | 0.23 (1.718)
  WBC count, Month 21, n=75: number analyzed (Participants) | 75
  WBC count, Month 21, n=75 | 0.30 (1.452)
  WBC count, Month 24, n=35: number analyzed (Participants) | 35
  WBC count, Month 24, n=35 | -0.04 (1.463)
  WBC count, Month 27, n=8: number analyzed (Participants) | 8
  WBC count, Month 27, n=8 | -0.05 (1.543)
  WBC count, Month 30, n=1: number analyzed (Participants) | 1
  WBC count, Month 30, n=1 | 0.40 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Basophil count, Month 15, n=99: number analyzed (Participants) | 99
  Basophil count, Month 15, n=99 | 0.009 (0.0292)
  Basophil count, Month 18, n=97: number analyzed (Participants) | 97
  Basophil count, Month 18, n=97 | 0.008 (0.0374)
  Basophil count, Month 21, n=75: number analyzed (Participants) | 75
  Basophil count, Month 21, n=75 | 0.001 (0.0243)
  Basophil count, Month 24, n=35: number analyzed (Participants) | 35
  Basophil count, Month 24, n=35 | -0.002 (0.0268)
  Basophil count, Month 27, n=8: number analyzed (Participants) | 8
  Basophil count, Month 27, n=8 | 0.010 (0.0351)
  Basophil count, Month 30, n=1: number analyzed (Participants) | 1
  Basophil count, Month 30, n=1 | 0.060 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Eosinophil count, Month 15, n=99: number analyzed (Participants) | 99
  Eosinophil count, Month 15, n=99 | 0.019 (0.1623)
  Eosinophil count, Month 18, n=97: number analyzed (Participants) | 97
  Eosinophil count, Month 18, n=97 | 0.008 (0.1609)
  Eosinophil count, Month 21, n=75: number analyzed (Participants) | 75
  Eosinophil count, Month 21, n=75 | -0.001 (0.1683)
  Eosinophil count, Month 24, n=35: number analyzed (Participants) | 35
  Eosinophil count, Month 24, n=35 | -0.033 (0.2489)
  Eosinophil count, Month 27, n=8: number analyzed (Participants) | 8
  Eosinophil count, Month 27, n=8 | -0.060 (0.0650)
  Eosinophil count, Month 30, n=1: number analyzed (Participants) | 1
  Eosinophil count, Month 30, n=1 | 0.010 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Lymphocyte count, Month 15, n=99: number analyzed (Participants) | 99
  Lymphocyte count, Month 15, n=99 | 0.1654 (0.53448)
  Lymphocyte count, Month 18, n=97: number analyzed (Participants) | 97
  Lymphocyte count, Month 18, n=97 | 0.1315 (0.71555)
  Lymphocyte count, Month 21, n=75: number analyzed (Participants) | 75
  Lymphocyte count, Month 21, n=75 | 0.0360 (0.51313)
  Lymphocyte count, Month 24, n=35: number analyzed (Participants) | 35
  Lymphocyte count, Month 24, n=35 | -0.1046 (0.50251)
  Lymphocyte count, Month 27, n=8: number analyzed (Participants) | 8
  Lymphocyte count, Month 27, n=8 | 0.0237 (0.47192)
  Lymphocyte count, Month 30, n=1: number analyzed (Participants) | 1
  Lymphocyte count, Month 30, n=1 | -0.2100 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Monocyte count, Month 15, n=99: number analyzed (Participants) | 99
  Monocyte count, Month 15, n=99 | 0.091 (0.1707)
  Monocyte count, Month 18, n=97: number analyzed (Participants) | 97
  Monocyte count, Month 18, n=97 | 0.085 (0.2257)
  Monocyte count, Month 21, n=75: number analyzed (Participants) | 75
  Monocyte count, Month 21, n=75 | 0.048 (0.1280)
  Monocyte count, Month 24, n=35: number analyzed (Participants) | 35
  Monocyte count, Month 24, n=35 | -0.009 (0.1228)
  Monocyte count, Month 27, n=8: number analyzed (Participants) | 8
  Monocyte count, Month 27, n=8 | -0.030 (0.1743)
  Monocyte count, Month 30, n=1: number analyzed (Participants) | 1
  Monocyte count, Month 30, n=1 | 0.110 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Neutrophil count, Month 15, n=99: number analyzed (Participants) | 99
  Neutrophil count, Month 15, n=99 | 0.365 (1.3448)
  Neutrophil count, Month 18, n=97: number analyzed (Participants) | 97
  Neutrophil count, Month 18, n=97 | -0.007 (1.2956)
  Neutrophil count, Month 21, n=75: number analyzed (Participants) | 75
  Neutrophil count, Month 21, n=75 | 0.211 (1.2534)
  Neutrophil count, Month 24, n=35: number analyzed (Participants) | 35
  Neutrophil count, Month 24, n=35 | 0.109 (1.2653)
  Neutrophil count, Month 27, n=8: number analyzed (Participants) | 8
  Neutrophil count, Month 27, n=8 | -0.003 (1.0602)
  Neutrophil count, Month 30, n=1: number analyzed (Participants) | 1
  Neutrophil count, Month 30, n=1 | 0.350 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

54. Secondary Outcome: Change From Baseline in Hematology Parameter-Red Blood Cell (RBC) Count From Month 15 to Month 30
Description: as for outcome 49
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
10^12 cells per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 0.17 (0.245)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | 0.19 (0.313)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 0.19 (0.248)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 0.16 (0.274)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 0.14 (0.267)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 0.10 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

55. Secondary Outcome: Change From Baseline in Hematology Parameter-Hemoglobin From Month 15 to Month 30
Description: as for outcome 50
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Grams per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | -0.71 (7.172)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | -0.29 (9.920)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | -1.09 (6.717)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | -2.26 (7.636)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | -3.25 (5.203)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | -4.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

56. Secondary Outcome: Change From Baseline in Hematology Parameter-Hematocrit From Month 15 to Month 30
Description: as for outcome 51
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Percentage of red blood cells in blood
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | -0.0133 (0.02272)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | -0.0134 (0.02963)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | -0.0091 (0.02346)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | -0.0102 (0.02364)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | -0.0166 (0.01935)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | -0.0340 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

57. Secondary Outcome: Change From Baseline in Hematology Parameter-Erythrocytes Mean Corpuscular Volume (MCV) From Month 15 to Month 30
Description: as for outcome 52
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Femtoliter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | -6.13 (2.724)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | -6.64 (3.004)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | -5.61 (3.413)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | -5.37 (2.691)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | -6.25 (3.770)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | -7.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

58. Secondary Outcome: Absolute Values of the Hematology Parameters: Platelet Count, WBC Count, Basophil Count, Eosinophil Count, Lymphocyte Count, Monocyte Count and Neutrophil Count
Description: Blood samples were collected for the analysis of hematology parameters including platelet count, WBC count, basophil count, eosinophil count, lymphocyte count, monocyte count and neutrophil count.
Time Frame: Up to Month 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
10^9 cells per liter
  Platelet count, n=100: number analyzed (Participants) | 100
  Platelet count, n=100 | 238.78 (56.321)
  WBC count, n=101: number analyzed (Participants) | 101
  WBC count, n=101 | 5.81 (1.606)
  Basophil count, n=101: number analyzed (Participants) | 101
  Basophil count, n=101 | 0.042 (0.0239)
  Eosinophil count, n=101: number analyzed (Participants) | 101
  Eosinophil count, n=101 | 0.160 (0.1305)
  Lymphocyte count, n=101: number analyzed (Participants) | 101
  Lymphocyte count, n=101 | 1.9528 (0.58037)
  Monocyte count, n=101: number analyzed (Participants) | 101
  Monocyte count, n=101 | 0.388 (0.1352)
  Neutrophil count, n=101: number analyzed (Participants) | 101
  Neutrophil count, n=101 | 3.269 (1.3055)

59. Secondary Outcome: Absolute Values of Hematology Parameter: RBC Count
Description: Blood samples were collected to analyze the hematology parameter: RBC count.
Time Frame: Up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
10^12 cells per liter | 4.84 (0.504)

60. Secondary Outcome: Absolute Values of Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin
Time Frame: Up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Grams per liter | 145.19 (11.121)

61. Secondary Outcome: Absolute Values of Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit (fraction of 1)
Time Frame: Up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Percentage of red blood cells in blood | 0.4445 (0.03412)

62. Secondary Outcome: Absolute Values of Hematology Parameter: Erythrocytes MCV
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes MCV.
Time Frame: Up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Femtoliter | 92.37 (5.546)

63. Secondary Outcome: Absolute Values of the Hematology Parameters of Platelet Count, WBC Count, Basophil Count, Eosinophil Count, Lymphocyte Count, Monocyte Count and Neutrophil Count From Month 15 to Month 30
Description: as for outcome 58
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
10^9 cells per Liter
  Platelet count, Month 15, n=99: number analyzed (Participants) | 99
  Platelet count, Month 15, n=99 | 245.56 (62.285)
  Platelet count, Month 18, n=97: number analyzed (Participants) | 97
  Platelet count, Month 18, n=97 | 250.99 (68.610)
  Platelet count, Month 21, n=75: number analyzed (Participants) | 75
  Platelet count, Month 21, n=75 | 247.04 (50.792)
  Platelet count, Month 24, n=35: number analyzed (Participants) | 35
  Platelet count, Month 24, n=35 | 245.43 (54.199)
  Platelet count, Month 27, n=8: number analyzed (Participants) | 8
  Platelet count, Month 27, n=8 | 271.63 (81.512)
  Platelet count, Month 30, n=1: number analyzed (Participants) | 1
  Platelet count, Month 30, n=1 | 417.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  WBC count, Month 15, n=99: number analyzed (Participants) | 99
  WBC count, Month 15, n=99 | 6.21 (1.983)
  WBC count, Month 18, n=97: number analyzed (Participants) | 97
  WBC count, Month 18, n=97 | 5.79 (1.748)
  WBC count, Month 21, n=75: number analyzed (Participants) | 75
  WBC count, Month 21, n=75 | 5.92 (1.626)
  WBC count, Month 24, n=35: number analyzed (Participants) | 35
  WBC count, Month 24, n=35 | 5.75 (1.377)
  WBC count, Month 27, n=8: number analyzed (Participants) | 8
  WBC count, Month 27, n=8 | 6.55 (1.787)
  WBC count, Month 30, n=1: number analyzed (Participants) | 1
  WBC count, Month 30, n=1 | 12.30 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Basophil count, Month 15, n=99: number analyzed (Participants) | 99
  Basophil count, Month 15, n=99 | 0.045 (0.0255)
  Basophil count, Month 18, n=97: number analyzed (Participants) | 97
  Basophil count, Month 18, n=97 | 0.044 (0.0344)
  Basophil count, Month 21, n=75: number analyzed (Participants) | 75
  Basophil count, Month 21, n=75 | 0.037 (0.0222)
  Basophil count, Month 24, n=35: number analyzed (Participants) | 35
  Basophil count, Month 24, n=35 | 0.033 (0.0214)
  Basophil count, Month 27, n=8: number analyzed (Participants) | 8
  Basophil count, Month 27, n=8 | 0.039 (0.0210)
  Basophil count, Month 30, n=1: number analyzed (Participants) | 1
  Basophil count, Month 30, n=1 | 0.090 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Eosinophil count, Month 15, n=99: number analyzed (Participants) | 99
  Eosinophil count, Month 15, n=99 | 0.163 (0.1238)
  Eosinophil count, Month 18, n=97: number analyzed (Participants) | 97
  Eosinophil count, Month 18, n=97 | 0.151 (0.1052)
  Eosinophil count, Month 21, n=75: number analyzed (Participants) | 75
  Eosinophil count, Month 21, n=75 | 0.141 (0.1085)
  Eosinophil count, Month 24, n=35: number analyzed (Participants) | 35
  Eosinophil count, Month 24, n=35 | 0.143 (0.1366)
  Eosinophil count, Month 27, n=8: number analyzed (Participants) | 8
  Eosinophil count, Month 27, n=8 | 0.090 (0.0366)
  Eosinophil count, Month 30, n=1: number analyzed (Participants) | 1
  Eosinophil count, Month 30, n=1 | 0.090 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Lymphocyte count, Month 15, n=99: number analyzed (Participants) | 99
  Lymphocyte count, Month 15, n=99 | 2.1271 (0.61543)
  Lymphocyte count, Month 18, n=97: number analyzed (Participants) | 97
  Lymphocyte count, Month 18, n=97 | 2.0999 (0.74371)
  Lymphocyte count, Month 21, n=75: number analyzed (Participants) | 75
  Lymphocyte count, Month 21, n=75 | 2.0521 (0.58855)
  Lymphocyte count, Month 24, n=35: number analyzed (Participants) | 35
  Lymphocyte count, Month 24, n=35 | 1.9229 (0.53307)
  Lymphocyte count, Month 27, n=8: number analyzed (Participants) | 8
  Lymphocyte count, Month 27, n=8 | 2.1350 (0.63370)
  Lymphocyte count, Month 30, n=1: number analyzed (Participants) | 1
  Lymphocyte count, Month 30, n=1 | 1.9100 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Monocyte count, Month 15, n=99: number analyzed (Participants) | 99
  Monocyte count, Month 15, n=99 | 0.451 (0.1617)
  Monocyte count, Month 18, n=97: number analyzed (Participants) | 97
  Monocyte count, Month 18, n=97 | 0.444 (0.2301)
  Monocyte count, Month 21, n=75: number analyzed (Participants) | 75
  Monocyte count, Month 21, n=75 | 0.423 (0.1379)
  Monocyte count, Month 24, n=35: number analyzed (Participants) | 35
  Monocyte count, Month 24, n=35 | 0.388 (0.0859)
  Monocyte count, Month 27, n=8: number analyzed (Participants) | 8
  Monocyte count, Month 27, n=8 | 0.396 (0.1640)
  Monocyte count, Month 30, n=1: number analyzed (Participants) | 1
  Monocyte count, Month 30, n=1 | 0.540 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Neutrophil count, Month 15, n=99: number analyzed (Participants) | 99
  Neutrophil count, Month 15, n=99 | 3.423 (1.6355)
  Neutrophil count, Month 18, n=97: number analyzed (Participants) | 97
  Neutrophil count, Month 18, n=97 | 3.056 (1.3502)
  Neutrophil count, Month 21, n=75: number analyzed (Participants) | 75
  Neutrophil count, Month 21, n=75 | 3.275 (1.2803)
  Neutrophil count, Month 24, n=35: number analyzed (Participants) | 35
  Neutrophil count, Month 24, n=35 | 3.273 (1.1311)
  Neutrophil count, Month 27, n=8: number analyzed (Participants) | 8
  Neutrophil count, Month 27, n=8 | 3.906 (1.6430)
  Neutrophil count, Month 30, n=1: number analyzed (Participants) | 1
  Neutrophil count, Month 30, n=1 | 9.640 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

64. Secondary Outcome: Absolute Values of Hematology Parameter-RBC Count From Month 15 to Month 30
Description: Blood samples were collected to analyze the hematology parameter: RBC count.
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
10^12 cells per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 4.85 (0.482)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | 4.85 (0.534)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 4.84 (0.474)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 4.90 (0.513)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 4.88 (0.557)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 5.10 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

65. Secondary Outcome: Absolute Values of Hematology Parameter-Hemoglobin From Month 15 to Month 30
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin.
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Grams per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 145.84 (10.827)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | 146.08 (14.021)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 144.52 (11.781)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 144.46 (11.559)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 138.25 (18.344)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 130.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

66. Secondary Outcome: Absolute Values of Hematology Parameter-Hematocrit From Month 15 to Month 30
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit (fraction of 1).
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Percentage of red blood cells in blood
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 0.4341 (0.03251)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | 0.4335 (0.04229)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 0.4349 (0.03472)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 0.4377 (0.03484)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 0.4183 (0.05263)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 0.3960 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

67. Secondary Outcome: Absolute Values of Hematology Parameter-Erythrocytes MCV From Month 15 to Month 30
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes MCV.
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Femtoliter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 90.16 (5.138)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | 89.64 (5.048)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 90.39 (5.533)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 89.74 (5.468)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 85.75 (4.652)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 78.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

68. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Parameters: Sodium, Potassium, Carbon-dioxide, Chloride, Glucose, Urea and Phosphate
Description: Blood samples were collected to analyze the chemistry parameters: Sodium, potassium, carbon dioxide, chloride, glucose, urea and phosphate. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Millimoles per liter
  Sodium | 0.2 (2.00)
  Potassium | 0.02 (0.295)
  Carbon dioxide | -0.0 (2.20)
  Chloride | -0.8 (2.34)
  Glucose | -0.37 (1.636)
  Urea | 0.13 (1.324)
  Phosphate | -0.005 (0.1853)

69. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: Creatinine and Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: Creatinine and Bilirubin. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Micromoles per liter
  Creatinine | -1.59 (14.736)
  Bilirubin | 0.9 (4.24)

70. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: ALT, ALP, AST, and Creatine Kinase
Description: Blood samples were collected to analyze the chemistry parameters: ALT, AST, ALP and creatine kinase. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
International units per liter
  ALT | 1.1 (14.17)
  AST | 0.5 (11.59)
  ALP | 0.3 (12.27)
  Creatine kinase | -29.1 (278.65)

71. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Glomerular Filtration Rate (GFR) From Creatinine Adjusted for Body Surface Area (BSA)
Description: Blood samples were collected from participants at indicated time points to analyze the clinical chemistry parameter: GFR from creatinine adjusted for BSA. Baseline is defined as the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline value is defined as post-dose value minus Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliters/seconds/1.73 meter square
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Milliliters/seconds/1.73 meter square | 0.00520 (0.221404)

72. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Lipase. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Units per liter | -2.3 (21.54)

73. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Albumin. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Grams per liter | 0.2 (2.54)

74. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Parameters: Sodium, Potassium, Carbon-dioxide, Chloride, Glucose, Urea and Phosphate From Month 15 to Month 30
Description: as for outcome 68
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Millimoles per liter
  Sodium, Month 15, n=99: number analyzed (Participants) | 99
  Sodium, Month 15, n=99 | -0.2 (1.93)
  Sodium, Month 18, n=97: number analyzed (Participants) | 97
  Sodium, Month 18, n=97 | -0.2 (1.78)
  Sodium, Month 21, n=75: number analyzed (Participants) | 75
  Sodium, Month 21, n=75 | -0.6 (1.97)
  Sodium, Month 24, n=35: number analyzed (Participants) | 35
  Sodium, Month 24, n=35 | -0.9 (2.39)
  Sodium, Month 27, n=8: number analyzed (Participants) | 8
  Sodium, Month 27, n=8 | -1.1 (2.03)
  Sodium, Month 30, n=1: number analyzed (Participants) | 1
  Sodium, Month 30, n=1 | -2.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Potassium, Month 15, n=99: number analyzed (Participants) | 99
  Potassium, Month 15, n=99 | 0.02 (0.325)
  Potassium, Month 18, n=97: number analyzed (Participants) | 97
  Potassium, Month 18, n=97 | 0.03 (0.315)
  Potassium, Month 21, n=75: number analyzed (Participants) | 75
  Potassium, Month 21, n=75 | -0.05 (0.321)
  Potassium, Month 24, n=35: number analyzed (Participants) | 35
  Potassium, Month 24, n=35 | -0.10 (0.335)
  Potassium, Month 27, n=8: number analyzed (Participants) | 8
  Potassium, Month 27, n=8 | -0.13 (0.271)
  Potassium, Month 30,n=1: number analyzed (Participants) | 1
  Potassium, Month 30,n=1 | 0.40 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Carbon dioxide, Month 15, n=99: number analyzed (Participants) | 99
  Carbon dioxide, Month 15, n=99 | 0.7 (2.10)
  Carbon dioxide, Month 18, n=97: number analyzed (Participants) | 97
  Carbon dioxide, Month 18, n=97 | 1.0 (2.26)
  Carbon dioxide, Month 21, n=75: number analyzed (Participants) | 75
  Carbon dioxide, Month 21, n=75 | 0.6 (1.86)
  Carbon dioxide, Month 24, n=35: number analyzed (Participants) | 35
  Carbon dioxide, Month 24, n=35 | 0.3 (2.09)
  Carbon dioxide, Month 27, n=8: number analyzed (Participants) | 8
  Carbon dioxide, Month 27, n=8 | 0.4 (2.72)
  Carbon dioxide, Month 30, n=1: number analyzed (Participants) | 1
  Carbon dioxide, Month 30, n=1 | 2.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Chloride, Month 15, n=99: number analyzed (Participants) | 99
  Chloride, Month 15, n=99 | -1.5 (2.29)
  Chloride, Month 18, n=97: number analyzed (Participants) | 97
  Chloride, Month 18, n=97 | -1.6 (2.31)
  Chloride, Month 21, n=75: number analyzed (Participants) | 75
  Chloride, Month 21, n=75 | -2.2 (2.30)
  Chloride, Month 24, n=35: number analyzed (Participants) | 35
  Chloride, Month 24, n=35 | -1.8 (2.21)
  Chloride, Month 27, n=8: number analyzed (Participants) | 8
  Chloride, Month 27, n=8 | -1.3 (1.58)
  Chloride, Month 30, n=1: number analyzed (Participants) | 1
  Chloride, Month 30, n=1 | -3.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Glucose, Month 15, n=99: number analyzed (Participants) | 99
  Glucose, Month 15, n=99 | 0.05 (1.907)
  Glucose, Month 18, n=97: number analyzed (Participants) | 97
  Glucose, Month 18, n=97 | 0.22 (2.804)
  Glucose, Month 21, n=75: number analyzed (Participants) | 75
  Glucose, Month 21, n=75 | 0.24 (2.033)
  Glucose, Month 24, n=35: number analyzed (Participants) | 35
  Glucose, Month 24, n=35 | 0.42 (2.546)
  Glucose, Month 27, n=8: number analyzed (Participants) | 8
  Glucose, Month 27, n=8 | -0.30 (1.278)
  Glucose, Month 30, n=1: number analyzed (Participants) | 1
  Glucose, Month 30, n=1 | -0.30 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Urea; Month 15, n=99: number analyzed (Participants) | 99
  Urea; Month 15, n=99 | -0.15 (1.157)
  Urea; Month 18, n=97: number analyzed (Participants) | 97
  Urea; Month 18, n=97 | 0.04 (1.364)
  Urea; Month 21, n=75: number analyzed (Participants) | 75
  Urea; Month 21, n=75 | -0.06 (1.271)
  Urea; Month 24, n=35: number analyzed (Participants) | 35
  Urea; Month 24, n=35 | 0.04 (1.114)
  Urea; Month 27 , n=8: number analyzed (Participants) | 8
  Urea; Month 27 , n=8 | 0.63 (1.458)
  Urea; Month 30, n=1: number analyzed (Participants) | 1
  Urea; Month 30, n=1 | 1.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Phosphate; Month 15, n=99: number analyzed (Participants) | 99
  Phosphate; Month 15, n=99 | 0.006 (0.2069)
  Phosphate; Month 18, n=97: number analyzed (Participants) | 97
  Phosphate; Month 18, n=97 | -0.007 (0.2015)
  Phosphate; Month 21, n=75: number analyzed (Participants) | 75
  Phosphate; Month 21, n=75 | 0.001 (0.1940)
  Phosphate; Month 24, n=35: number analyzed (Participants) | 35
  Phosphate; Month 24, n=35 | -0.009 (0.2248)
  Phosphate; Month 27, n=8: number analyzed (Participants) | 8
  Phosphate; Month 27, n=8 | 0.031 (0.2120)
  Phosphate; Month 30, n=1: number analyzed (Participants) | 1
  Phosphate; Month 30, n=1 | 0.350 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

75. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: Creatinine and Bilirubin From Month 15 to Month 30
Description: as for outcome 69
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Micromoles per liter
  Creatinine, Month 15, n=99: number analyzed (Participants) | 99
  Creatinine, Month 15, n=99 | -2.73 (13.479)
  Creatinine, Month 18, n=97: number analyzed (Participants) | 97
  Creatinine, Month 18, n=97 | 3.19 (12.588)
  Creatinine, Month 21, n=75: number analyzed (Participants) | 75
  Creatinine, Month 21, n=75 | -2.92 (14.496)
  Creatinine, Month 24, n=35: number analyzed (Participants) | 35
  Creatinine, Month 24, n=35 | -6.80 (16.452)
  Creatinine, Month 27, n=8: number analyzed (Participants) | 8
  Creatinine, Month 27, n=8 | -6.95 (9.095)
  Creatinine, Month 30, n=1: number analyzed (Participants) | 1
  Creatinine, Month 30, n=1 | -10.60 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Bilirubin, Month 15, n=99: number analyzed (Participants) | 99
  Bilirubin, Month 15, n=99 | 0.7 (4.99)
  Bilirubin, Month 18, n=97: number analyzed (Participants) | 97
  Bilirubin, Month 18, n=97 | 0.4 (4.42)
  Bilirubin, Month 21 n=75: number analyzed (Participants) | 75
  Bilirubin, Month 21 n=75 | 1.7 (4.34)
  Bilirubin, Month 24, n=35: number analyzed (Participants) | 35
  Bilirubin, Month 24, n=35 | 1.9 (5.75)
  Bilirubin, Month 27 n=8: number analyzed (Participants) | 8
  Bilirubin, Month 27 n=8 | 0.8 (1.04)
  Bilirubin, Month 30, n=1: number analyzed (Participants) | 1
  Bilirubin, Month 30, n=1 | -4.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

76. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: ALT, ALP, AST, and Creatine Kinase From Month 15 to Month 30
Description: as for outcome 70
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
International units per liter
  ALT, Month 15, n=99: number analyzed (Participants) | 99
  ALT, Month 15, n=99 | 4.0 (20.92)
  ALT, Month 18, n=97: number analyzed (Participants) | 97
  ALT, Month 18, n=97 | 2.9 (14.96)
  ALT, Month 21, n=75: number analyzed (Participants) | 75
  ALT, Month 21, n=75 | 3.1 (23.81)
  ALT, Month 24, n=35: number analyzed (Participants) | 35
  ALT, Month 24, n=35 | -0.2 (12.35)
  ALT, Month 27, n=8: number analyzed (Participants) | 8
  ALT, Month 27, n=8 | 1.6 (16.16)
  ALT, Month 30 n=1: number analyzed (Participants) | 1
  ALT, Month 30 n=1 | -2.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  ALP, Month 15, n=99: number analyzed (Participants) | 99
  ALP, Month 15, n=99 | -2.1 (13.62)
  ALP, Month 18, n=97: number analyzed (Participants) | 97
  ALP, Month 18, n=97 | -0.8 (14.45)
  ALP, Month 21, n=75: number analyzed (Participants) | 75
  ALP, Month 21, n=75 | -0.2 (13.61)
  ALP, Month 24, n=35: number analyzed (Participants) | 35
  ALP, Month 24, n=35 | 0.1 (10.35)
  ALP, Month 27, n=8: number analyzed (Participants) | 8
  ALP, Month 27, n=8 | 5.5 (12.32)
  ALP, Month 30, n=1: number analyzed (Participants) | 1
  ALP, Month 30, n=1 | -9.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  AST, Month 15, n=99: number analyzed (Participants) | 99
  AST, Month 15, n=99 | 1.2 (9.63)
  AST, Month 18, n=97: number analyzed (Participants) | 97
  AST, Month 18, n=97 | 4.1 (26.52)
  AST, Month 21, n=75: number analyzed (Participants) | 75
  AST, Month 21, n=75 | 1.4 (8.80)
  AST, Month 24, n=35: number analyzed (Participants) | 35
  AST, Month 24, n=35 | -0.5 (5.54)
  AST, Month 27, n=8: number analyzed (Participants) | 8
  AST, Month 27, n=8 | 1.6 (9.65)
  AST, Month 30, n=1: number analyzed (Participants) | 1
  AST, Month 30, n=1 | -1.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Creatine Kinase, Month 15, n=99: number analyzed (Participants) | 99
  Creatine Kinase, Month 15, n=99 | -25.0 (306.57)
  Creatine Kinase, Month 18, n=97: number analyzed (Participants) | 97
  Creatine Kinase, Month 18, n=97 | 132.5 (1053.02)
  Creatine Kinase, Month 21, n=75: number analyzed (Participants) | 75
  Creatine Kinase, Month 21, n=75 | 28.0 (454.78)
  Creatine Kinase, Month 24, n=35: number analyzed (Participants) | 35
  Creatine Kinase, Month 24, n=35 | -61.7 (376.27)
  Creatine Kinase, Month 27, n=8: number analyzed (Participants) | 8
  Creatine Kinase, Month 27, n=8 | 70.8 (107.32)
  Creatine Kinase, Month 30, n=1: number analyzed (Participants) | 1
  Creatine Kinase, Month 30, n=1 | -8.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

77. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter-glomerular Filtration Rate (GFR) From Creatinine Adjusted for Body Surface Area (BSA) From Month 15 to Month 30
Description: as for outcome 71
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Milliliters/seconds/1.73 meter square
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Milliliters/seconds/1.73 meter square
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 0.03216 (0.210193)
  Month 18, n=93: number analyzed (Participants) | 93
  Month 18, n=93 | -0.09140 (0.190551)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 0.02044 (0.203936)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 0.07667 (0.252677)
  Month 27, n=7: number analyzed (Participants) | 7
  Month 27, n=7 | 0.06905 (0.173056)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 0.20000 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

78. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter- Lipase From Month 15 to Month 30
Description: as for outcome 72
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Units per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 2.2 (32.47)
  Month 18, n=93: number analyzed (Participants) | 93
  Month 18, n=93 | 0.9 (31.03)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | -1.3 (29.74)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | -9.9 (53.42)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 5.9 (23.43)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 2.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

79. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter-Albumin From Month 15 to Month 30
Description: Blood samples were collected for the analysis of clinical chemistry parameter-Albumin. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Grams per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | -0.0 (2.63)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | -0.2 (2.75)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | -0.3 (2.16)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | -0.5 (2.09)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 0.0 (1.85)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 0.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

80. Secondary Outcome: Absolute Values of Clinical Chemistry Laboratory Parameters: Sodium, Potassium, Carbon-dioxide, Chloride, Glucose, Urea and Phosphate
Description: Blood samples were collected to analyze the chemistry parameters: Sodium, potassium, carbon dioxide, chloride, glucose, urea and phosphate.
Time Frame: Up to Month 12
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Millimoles per liter
  Sodium | 139.7 (1.67)
  Potassium | 4.15 (0.309)
  Carbon dioxide | 23.1 (2.02)
  Chloride | 103.8 (2.18)
  Glucose | 5.26 (1.425)
  Urea | 5.08 (1.588)
  Phosphate | 1.087 (0.1687)

81. Secondary Outcome: Absolute Values of Clinical Laboratory Parameters: Creatinine and Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: Creatinine and Bilirubin.
Time Frame: Up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Micromoles per liter
  Creatinine | 89.10 (15.229)
  Bilirubin | 10.0 (5.10)

82. Secondary Outcome: Absolute Values of Clinical Laboratory Parameters: ALT, ALP, AST, and Creatine Kinase
Description: Blood samples were collected to analyze the chemistry parameters: ALT, AST, ALP and creatine kinase.
Time Frame: Up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
International units per liter
  ALT | 24.6 (17.52)
  AST | 21.7 (14.31)
  ALP | 69.0 (19.42)
  Creatine kinase | 181.4 (153.58)

83. Secondary Outcome: Absolute Values of Clinical Laboratory Parameter: Glomerular Filtration Rate (GFR) From Creatinine Adjusted for Body Surface Area (BSA)
Description: Blood samples were collected from participants to analyze the clinical chemistry parameter: GFR from Creatinine adjusted for BSA
Time Frame: Up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliters/seconds/1.73 meter square
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Milliliters/seconds/1.73 meter square | 1.60853 (0.305979)

84. Secondary Outcome: Absolute Values of Clinical Laboratory Parameter: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Lipase.
Time Frame: Up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Units per liter | 31.6 (25.92)

85. Secondary Outcome: Absolute Values of Clinical Laboratory Parameter: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Albumin.
Time Frame: Up to Month 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 101
Grams per liter | 44.7 (2.74)

86. Secondary Outcome: Absolute Values of Clinical Chemistry Laboratory Parameters of Sodium, Potassium, Carbon-dioxide, Chloride, Glucose, Urea and Phosphate From Month 15 to Month 30
Description: as for outcome 80
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Millimoles per liter
  Sodium, Month 15, n=99: number analyzed (Participants) | 99
  Sodium, Month 15, n=99 | 139.3 (1.81)
  Sodium, Month 18, n=97: number analyzed (Participants) | 97
  Sodium, Month 18, n=97 | 139.3 (1.92)
  Sodium, Month 21, n=75: number analyzed (Participants) | 75
  Sodium, Month 21, n=75 | 139.0 (1.89)
  Sodium, Month 24, n=35: number analyzed (Participants) | 35
  Sodium, Month 24, n=35 | 138.7 (1.87)
  Sodium, Month 27, n=8: number analyzed (Participants) | 8
  Sodium, Month 27, n=8 | 138.1 (1.36)
  Sodium, Month 30, n=1: number analyzed (Participants) | 1
  Sodium, Month 30, n=1 | 137.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Potassium, Month 15, n=99: number analyzed (Participants) | 99
  Potassium, Month 15, n=99 | 4.15 (0.366)
  Potassium, Month 18, n=97: number analyzed (Participants) | 97
  Potassium, Month 18, n=97 | 4.16 (0.340)
  Potassium, Month 21, n=75: number analyzed (Participants) | 75
  Potassium, Month 21, n=75 | 4.08 (0.313)
  Potassium, Month 24, n=35: number analyzed (Participants) | 35
  Potassium, Month 24, n=35 | 4.02 (0.308)
  Potassium, Month 27, n=8: number analyzed (Participants) | 8
  Potassium, Month 27, n=8 | 3.94 (0.119)
  Potassium, Month 30,n=1: number analyzed (Participants) | 1
  Potassium, Month 30,n=1 | 4.10 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Carbon dioxide, Month 15, n=99: number analyzed (Participants) | 99
  Carbon dioxide, Month 15, n=99 | 23.8 (2.18)
  Carbon dioxide, Month 18, n=97: number analyzed (Participants) | 97
  Carbon dioxide, Month 18, n=97 | 24.1 (2.11)
  Carbon dioxide, Month 21, n=75: number analyzed (Participants) | 75
  Carbon dioxide, Month 21, n=75 | 23.8 (2.24)
  Carbon dioxide, Month 24, n=35: number analyzed (Participants) | 35
  Carbon dioxide, Month 24, n=35 | 23.8 (2.09)
  Carbon dioxide, Month 27, n=8: number analyzed (Participants) | 8
  Carbon dioxide, Month 27, n=8 | 23.5 (2.27)
  Carbon dioxide, Month 30, n=1: number analyzed (Participants) | 1
  Carbon dioxide, Month 30, n=1 | 24.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Chloride, Month 15, n=99: number analyzed (Participants) | 99
  Chloride, Month 15, n=99 | 103.1 (2.29)
  Chloride, Month 18, n=97: number analyzed (Participants) | 97
  Chloride, Month 18, n=97 | 103.0 (2.37)
  Chloride, Month 21, n=75: number analyzed (Participants) | 75
  Chloride, Month 21, n=75 | 102.6 (2.24)
  Chloride, Month 24, n=35: number analyzed (Participants) | 35
  Chloride, Month 24, n=35 | 102.9 (2.18)
  Chloride, Month 27, n=8: number analyzed (Participants) | 8
  Chloride, Month 27, n=8 | 103.0 (1.85)
  Chloride, Month 30, n=1: number analyzed (Participants) | 1
  Chloride, Month 30, n=1 | 101.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Glucose, Month 15, n=99: number analyzed (Participants) | 99
  Glucose, Month 15, n=99 | 5.72 (2.344)
  Glucose, Month 18, n=97: number analyzed (Participants) | 97
  Glucose, Month 18, n=97 | 5.89 (3.089)
  Glucose, Month 21, n=75: number analyzed (Participants) | 75
  Glucose, Month 21, n=75 | 5.86 (2.382)
  Glucose, Month 24, n=35: number analyzed (Participants) | 35
  Glucose, Month 24, n=35 | 6.14 (3.294)
  Glucose, Month 27, n=8: number analyzed (Participants) | 8
  Glucose, Month 27, n=8 | 5.33 (0.654)
  Glucose, Month 30, n=1: number analyzed (Participants) | 1
  Glucose, Month 30, n=1 | 4.40 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Urea; Month 15, n=99: number analyzed (Participants) | 99
  Urea; Month 15, n=99 | 4.81 (1.362)
  Urea; Month 18, n=97: number analyzed (Participants) | 97
  Urea; Month 18, n=97 | 4.96 (1.413)
  Urea; Month 21, n=75: number analyzed (Participants) | 75
  Urea; Month 21, n=75 | 4.94 (1.529)
  Urea; Month 24, n=35: number analyzed (Participants) | 35
  Urea; Month 24, n=35 | 4.79 (1.313)
  Urea; Month 27 , n=8: number analyzed (Participants) | 8
  Urea; Month 27 , n=8 | 5.69 (1.668)
  Urea; Month 30, n=1: number analyzed (Participants) | 1
  Urea; Month 30, n=1 | 5.00 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Phosphate; Month 15, n=99: number analyzed (Participants) | 99
  Phosphate; Month 15, n=99 | 1.091 (0.1919)
  Phosphate; Month 18, n=97: number analyzed (Participants) | 97
  Phosphate; Month 18, n=97 | 1.079 (0.1844)
  Phosphate; Month 21, n=75: number analyzed (Participants) | 75
  Phosphate; Month 21, n=75 | 1.083 (0.1848)
  Phosphate; Month 24, n=35: number analyzed (Participants) | 35
  Phosphate; Month 24, n=35 | 1.091 (0.1574)
  Phosphate; Month 27, n=8: number analyzed (Participants) | 8
  Phosphate; Month 27, n=8 | 1.119 (0.1252)
  Phosphate; Month 30, n=1: number analyzed (Participants) | 1
  Phosphate; Month 30, n=1 | 1.300 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

87. Secondary Outcome: Absolute Values of Clinical Laboratory Parameters: Creatinine and Bilirubin From Month 15 to Month 30
Description: Blood samples were collected to analyze the chemistry parameters: Creatinine and Bilirubin.
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Micromoles per liter
  Creatinine, Month 15, n=99: number analyzed (Participants) | 99
  Creatinine, Month 15, n=99 | 88.50 (13.908)
  Creatinine, Month 18, n=97: number analyzed (Participants) | 97
  Creatinine, Month 18, n=97 | 94.26 (12.797)
  Creatinine, Month 21, n=75: number analyzed (Participants) | 75
  Creatinine, Month 21, n=75 | 88.09 (14.410)
  Creatinine, Month 24, n=35: number analyzed (Participants) | 35
  Creatinine, Month 24, n=35 | 87.77 (14.390)
  Creatinine, Month 27, n=8: number analyzed (Participants) | 8
  Creatinine, Month 27, n=8 | 88.85 (12.854)
  Creatinine, Month 30, n=1: number analyzed (Participants) | 1
  Creatinine, Month 30, n=1 | 91.90 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Bilirubin, Month 15, n=99: number analyzed (Participants) | 99
  Bilirubin, Month 15, n=99 | 9.9 (4.67)
  Bilirubin, Month 18, n=97: number analyzed (Participants) | 97
  Bilirubin, Month 18, n=97 | 9.5 (4.69)
  Bilirubin, Month 21 n=75: number analyzed (Participants) | 75
  Bilirubin, Month 21 n=75 | 10.7 (5.49)
  Bilirubin, Month 24, n=35: number analyzed (Participants) | 35
  Bilirubin, Month 24, n=35 | 10.9 (6.69)
  Bilirubin, Month 27 n=8: number analyzed (Participants) | 8
  Bilirubin, Month 27 n=8 | 8.5 (4.38)
  Bilirubin, Month 30, n=1: number analyzed (Participants) | 1
  Bilirubin, Month 30, n=1 | 4.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

88. Secondary Outcome: Absolute Values of Clinical Laboratory Parameters: ALT, ALP, AST, and Creatine Kinase From Month 15 to Month 30
Description: Blood samples were collected to analyze the chemistry parameters: ALT, AST, ALP and creatine kinase.
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
International units per liter
  ALT, Month 15, n=99: number analyzed (Participants) | 99
  ALT, Month 15, n=99 | 27.9 (23.06)
  ALT, Month 18, n=97: number analyzed (Participants) | 97
  ALT, Month 18, n=97 | 26.4 (16.91)
  ALT, Month 21, n=75: number analyzed (Participants) | 75
  ALT, Month 21, n=75 | 26.2 (23.02)
  ALT, Month 24, n=35: number analyzed (Participants) | 35
  ALT, Month 24, n=35 | 24.1 (12.23)
  ALT, Month 27, n=8: number analyzed (Participants) | 8
  ALT, Month 27, n=8 | 24.1 (8.03)
  ALT, Month 30 n=1: number analyzed (Participants) | 1
  ALT, Month 30 n=1 | 17.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  ALP, Month 15, n=99: number analyzed (Participants) | 99
  ALP, Month 15, n=99 | 66.3 (19.77)
  ALP, Month 18, n=97: number analyzed (Participants) | 97
  ALP, Month 18, n=97 | 67.5 (22.26)
  ALP, Month 21, n=75: number analyzed (Participants) | 75
  ALP, Month 21, n=75 | 68.3 (21.10)
  ALP, Month 24, n=35: number analyzed (Participants) | 35
  ALP, Month 24, n=35 | 65.9 (18.86)
  ALP, Month 27, n=8: number analyzed (Participants) | 8
  ALP, Month 27, n=8 | 76.9 (15.25)
  ALP, Month 30, n=1: number analyzed (Participants) | 1
  ALP, Month 30, n=1 | 70.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  AST, Month 15, n=99: number analyzed (Participants) | 99
  AST, Month 15, n=99 | 22.4 (10.72)
  AST, Month 18, n=97: number analyzed (Participants) | 97
  AST, Month 18, n=97 | 25.2 (27.55)
  AST, Month 21, n=75: number analyzed (Participants) | 75
  AST, Month 21, n=75 | 21.7 (8.73)
  AST, Month 24, n=35: number analyzed (Participants) | 35
  AST, Month 24, n=35 | 19.8 (5.57)
  AST, Month 27, n=8: number analyzed (Participants) | 8
  AST, Month 27, n=8 | 20.5 (5.32)
  AST, Month 30, n=1: number analyzed (Participants) | 1
  AST, Month 30, n=1 | 14.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Creatine Kinase, Month 15, n=99: number analyzed (Participants) | 99
  Creatine Kinase, Month 15, n=99 | 178.6 (198.96)
  Creatine Kinase, Month 18, n=97: number analyzed (Participants) | 97
  Creatine Kinase, Month 18, n=97 | 338.4 (1050.63)
  Creatine Kinase, Month 21, n=75: number analyzed (Participants) | 75
  Creatine Kinase, Month 21, n=75 | 226.9 (374.26)
  Creatine Kinase, Month 24, n=35: number analyzed (Participants) | 35
  Creatine Kinase, Month 24, n=35 | 151.9 (70.67)
  Creatine Kinase, Month 27, n=8: number analyzed (Participants) | 8
  Creatine Kinase, Month 27, n=8 | 251.9 (139.79)
  Creatine Kinase, Month 30, n=1: number analyzed (Participants) | 1
  Creatine Kinase, Month 30, n=1 | 165.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

89. Secondary Outcome: Absolute Values of Clinical Laboratory Parameter-glomerular Filtration Rate (GFR) From Creatinine Adjusted for Body Surface Area (BSA) From Month 15 to Month 30
Description: as for outcome 83
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Milliliters/seconds/1.73 meter square
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Milliliters/seconds/1.73 meter square
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 1.62074 (0.285224)
  Month 18, n=93: number analyzed (Participants) | 93
  Month 18, n=93 | 1.51293 (0.275550)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 1.58759 (0.293326)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 1.61813 (0.292292)
  Month 27, n=7: number analyzed (Participants) | 7
  Month 27, n=7 | 1.68813 (0.187510)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 1.81670 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

90. Secondary Outcome: Absolute Values of Clinical Laboratory Parameter-Lipase From Month 15 to Month 30
Description: Blood samples were collected for the analysis of clinical chemistry parameter-Lipase.
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Units per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 36.0 (33.52)
  Month 18, n=93: number analyzed (Participants) | 93
  Month 18, n=93 | 35.0 (30.44)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 34.5 (33.39)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 34.6 (26.30)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 38.6 (30.26)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 35.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

91. Secondary Outcome: Absolute Values of Clinical Laboratory Parameter-Albumin From Month 15 to Month 30
Description: Blood samples were collected for the analysis of clinical chemistry parameter-Albumin.
Time Frame: Months 15, 18, 21, 24, 27, 30
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 115
Grams per liter
  Month 15, n=99: number analyzed (Participants) | 99
  Month 15, n=99 | 44.5 (3.02)
  Month 18, n=97: number analyzed (Participants) | 97
  Month 18, n=97 | 44.3 (2.71)
  Month 21, n=75: number analyzed (Participants) | 75
  Month 21, n=75 | 44.1 (2.49)
  Month 24, n=35: number analyzed (Participants) | 35
  Month 24, n=35 | 43.7 (3.05)
  Month 27, n=8: number analyzed (Participants) | 8
  Month 27, n=8 | 43.8 (2.82)
  Month 30, n=1: number analyzed (Participants) | 1
  Month 30, n=1 | 39.0 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

92. Other Pre Specified Outcome: Change From Baseline in Urinalysis Parameters: Urine Albumin to Creatinine Ratio
Description: Urine samples were not planned to be collected for the analysis of urine albumin to creatinine ratio. The results for this outcome measure will never be posted.
Time Frame: Baseline and up to Month 12
Population: Safety population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 0

93. Other Pre Specified Outcome: Change From Baseline in Urinalysis Parameters: Urine Protein to Creatinine Ratio
Description: Urine samples were not planned to be collected for the analysis of urine protein to creatinine ratio. The results for this outcome measure will never be posted.
Time Frame: Baseline and up to Month 12
Population: as for outcome 92
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 0

94. Other Pre Specified Outcome: Change From Baseline in Urinalysis Parameters: Urine Phosphate
Description: Urine samples were not planned to be collected for the analysis of urine phosphate. The results for this outcome measure will never be posted.
Time Frame: Baseline and up to Month 12
Population: as for outcome 92
Arm/Group | Participants With HIV Infection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs), non-serious AEs and all-cause mortality were collected up to 30 months
Description: Adverse events were reported for Safety Population which comprised of all participants enrolled,who received atleast 1 dose of CAB LA+RPV LA.Study staff participants only provided input through completion of surveys,semi-structured interviews and facilitation calls and didn't have to complete the informed consent process and did not receive oral lead-in medication or CAB+RPV LA injections. Adverse events for study staff participants were not collected because it was not required per study design
Arm/Group | Participants With HIV Infection
All-Cause Mortality (participants affected / at risk) | 1/115
Serious Adverse Events (participants affected / at risk) | 9/115
Other Adverse Events (participants affected / at risk) | 101/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With HIV Infection (N=115)
Mental status changes (Psychiatric disorders) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With HIV Infection (N=115)
Injection site pain (General disorders) | 64 (720)
Injection site discomfort (General disorders) | 30 (259)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (25)
Diarrhoea (Gastrointestinal disorders) | 20 (23)
Fatigue (General disorders) | 23 (53)
Injection site induration (General disorders) | 15 (27)
Headache (Nervous system disorders) | 16 (26)
Injection site nodule (General disorders) | 14 (25)
Injection site swelling (General disorders) | 14 (27)
Insomnia (Psychiatric disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 13 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Injection site bruising (General disorders) | 10 (13)
Rash (Skin and subcutaneous tissue disorders) | 10 (12)
COVID-19 (Infections and infestations) | 18 (18)
Influenza (Infections and infestations) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (16)
Proctitis gonococcal (Infections and infestations) | 7 (8)
Pyrexia (General disorders) | 9 (28)
Sinusitis (Infections and infestations) | 8 (8)
Chills (General disorders) | 7 (8)
Nasopharyngitis (Infections and infestations) | 11 (11)
Syphilis (Infections and infestations) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 9 (12)
Oropharyngeal gonococcal infection (Infections and infestations) | 8 (10)
Pharyngitis (Infections and infestations) | 8 (11)
Gastroenteritis (Infections and infestations) | 7 (9)
Pharyngitis streptococcal (Infections and infestations) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Depression (Psychiatric disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 6 (6)
Dysuria (Renal and urinary disorders) | 7 (7)
Blood creatine phosphokinase increased (Investigations) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT04001803/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT04001803/SAP_002.pdf